# Cover Page for ClinicalTrials.gov

# **Document:**

Study Protocol

PI: Ronald Cohen

# **Official Study Title:**

The WISE (Weightloss Intervention Surgical Effects) Brain Study (WISEBrain)

**NCT#:** NCT02137070

Document Date: January 20, 2022

# **Protocol**

 Project Title: Obesity and Type 2 Diabetes; Bariatric Surgery Effects on Brain Function

**Short Title:** WISE Brain Function Study (Weight Loss Intervention and Surgical Effects on Brain Function.)

2. Primary Investigator: Ron A. Cohen, Ph.D., ABPP, ABCN

**<u>Co-Investigators:</u>** Kenneth Cusi, M.D.

Michael Marsiske, Ph.D. Adam J. Woods, Ph.D.

Song Lai, Ph.D.

Christiaan Leeuwenburgh, Ph.D.

Steve Anton, Ph.D. Jeffrey Friedman, M.D.

Yenisel Cruz-Almeida, M.S.P.H., Ph.D.

Eric Porges, Ph.D.

Stephan Eisenschenk, M.D.

Source of Funding: NIDKK- NIH

# 3. Abstract:

It is important to highlight the fact that the bariatric surgery intervention itself is NOT a part of this research protocol. The UFHealth Shands Bariatric Surgical Team is operating independently of this study, with regard to decisions involving the suitability of candidates for bariatric surgery. The research team is not involved in any of those patient and physician decisions. Once patients have decided to move forward with bariatric surgery, they will be provided information on the WISE Brain Study, and be given an option of participating in research that will run in parallel to their surgical intervention. This study is designed to examine the effects of the bariatric surgery and resultant weight loss on cognition.

The proposed study will delineate mechanisms underlying the effect of chronic obesity on brain functioning and determine if cognitive benefits of bariatric surgery and weight loss contribute to enhanced cerebral metabolic or hemodynamic function assessed using multimodal neuroimaging methods. The contribution of post-surgical improvements in diabetes-associated insulin-glucose disturbances will be tested. Obesity has reached epidemic proportions and is now a major public health problem, contributing to various comorbid medical conditions, including brain disturbances. There is increasing evidence that chronic obesity may adversely affect the brain, even in the absence of comorbid diseases, such as diabetes, cardiovascular disease, and stroke. We have previously shown that elevated body mass index (BMI) is associated with reduced cognitive function. Increasingly, bariatric surgery is being used as a

treatment for chronic morbid obesity. Besides causing dramatic weight loss in many patients, bariatric surgery alters systemic metabolic and vascular function, including altering insulin and glucose metabolism. Our initial findings from a multicenter longitudinal study of bariatric surgery indicated that people experience improvements in neurocognitive functioning, including memory recall, by 12 weeks post-surgery. These benefits continue over 12 months and relate to not only the amount of weight lost, but also changes in underlying risk factors, such as improved metabolic function, and remission of type-2 diabetes. Neuroimaging provides a potentially powerful biomarker of alterations in brain structure and function (e.g., FMRI), as well as cerebral pathophysiology. To date, no published studies have examined neuronal, metabolic and vascular brain changes following bariatric surgery as proposed in this study. Our preliminary neuroimaging data indicates enhanced functional brain response on FMRI, increased regional cerebral blood flow on arterial spin labeling (ASL), and changes in cerebral metabolite levels on magnetic resonance spectroscopy (MRS). We hypothesize that: 1) Cerebral metabolic and hemodynamic disturbances linked to obesity adversely affect brain function (evident from cognitive testing and FMRI); 2) Weight loss and associated metabolic changes post-bariatric surgery improve brain functions; and 3) Enhanced neurocognitive and neuronal function (FMRI) are due to improved cerebral metabolic (MRS) and vascular (ASL) function. Remission of diabetes is expected to be one factor accounting for these effects, though this effect will also be tied to improved cerebral (MRS) and systemic (e.g., serum cytokines) metabolic health and cerebral perfusion (ASL). A prospective longitudinal cohort matched design will be used to assess changes in these neuroimaging indices, pre- and postsurgery and relative non-surgical obese controls. The groups will have equal proportions of diabetics and non-diabetics with obesity, enabling us to test its influence. By examining obesity and weight loss in the context of bariatric surgery, this study capitalizes on a powerful natural experimental manipulation that can provide a unique window into the effects of obesity and weight loss on the brain.

# 4. Background:

There is mounting evidence that severe obesity is a risk factor for brain dysfunction. This study examines the effects of obesity on the brain but moves beyond previous research by employing an experimental design to delineate the effects of weight loss following bariatric surgery on brain function and underlying pathophysiology. The proposed study has compelling scientific, clinical, and public health significance.

**Public health/clinical significance**: **1)** Obesity is a major public health problem contributing to various medical problems that affect mortality and morbidity  $^{26}$ ; **2)** Currently, over 15 million Americans (1 in 20) are severely obese, and the prevalence of severe obesity is accelerating  $^{27}$ . Severe obesity has major public health and socioeconomic consequences, including increasing health care expenditures  $^{2}$ , and reducing productivity  $^{28}$   $^{29}$  and quality of life (QOL)  $^{30}$ ; **3)** Severely obese people often experience neurocognitive impairments that further diminish health status, health care behavior and utilization, treatment adherence, and QOL; **4)** No study has used neuroimaging approaches to examine whether dramatic weight

loss via bariatric surgery produces changes in obesity-related brain dysfunction; **5)** Evidence of improved brain function post-surgically would motivate future dose-response research to determine whether benefits are achieved from more modest weight loss through behavioral and pharmacological treatments; **6)** Biomarkers of obesity-related brain disturbance may be identified that may inform and enhance future clinical practice, providing additional rationale for aggressively treating obesity in people at risk for brain dysfunction; **7)** Evidence of obesity-associated brain dysfunction may signal a need for interventions to ensure adherence to post-operative behavioral demands.

Adult obesity is highly prevalent and affects health as people age. Millions of obese Americans are now in middle age, a period of life when risk for more serious medical problems increases significantly  $^{31-33}$ . Obesity affects over 40% of these adults, and severe obesity [body mass index (BMI)  $\geq$  40 kg/m $^2$ ] is increasing at twice the rate of moderate obesity  $^{27}$ . Severely obese adults have increased risk for co-morbidities, with over 75% developing one or more comorbidities (e.g., diabetes, hypertension, arthritis) with advanced age  $^{27,34-41}$ . Cognitive dysfunction affects health status, QOL, and treatment adherence. Brain dysfunction occurs secondary to illness that increases mortality, and it adversely affects health status  $^{42-46}$ . Even mild cognitive deficits affect QOL, diet, physical activity, and other health behaviors  $^{45,47-49}$ , and they are often found to be a stronger predictor of health outcome than other clinical factors  $^{42}$ , but they typically receive less clinical attention.

Obesity-associated metabolic and vascular disturbances contribute to brain dysfunction. Diabetes and vascular disease are among the most common conditions resulting from severe obesity 50-60. It is now well-established that chronic diabetes and vascular disease contribute to brain dysfunction 19,20,61-68 25,58-60,69-71. These effects occur even in the absence of large vessel stroke 19,62,65,67, increasing the risk for dementia later in life 14-15,18-20,22. Accordingly, obesity-associated brain dysfunction has major public health implications as the U.S. population ages and the obesity epidemic continues. This provides a strong rationale for the proposed study.

Cognitive dysfunction affects medical and surgical outcome <sup>42,43,72</sup>. Furthermore, people with cognitive deficits lose less weight following bariatric surgery (see preliminary data; section C.10).

Obesity is a modifiable risk factor for cognitive decline and diminished brain health. Weight reduction has been shown to improve health status and reduce disease risk 73-75. Our past studies indicate that cognitive functions also improves with weight loss following bariatric surgery (see preliminary data) 17,18,76.

Bariatric surgery is effective and increasingly popular. The prevalence and refractoriness of severe obesity led to bariatric surgery becoming an established treatment for severe obesity  $^{77}$ . Bariatric surgeries in the U.S. increased over 14-fold (from 13,386 to > 210,000) from 1998 to 2010  $^{78}$ . The surgery is an effective method for rapidly producing significant weight loss,

<sup>79-81</sup>, as most severely obese patients lose 50% to 75% of their excess weight within two years post-surgery, with many maintaining this weight loss for 10 years or longer <sup>81-86</sup>. Partial or total resolution of comorbidities, including diabetes, tends to occur, along with reductions in mortality. <sup>81,82,84-87</sup>. It may also be cost-effective relative to life-long pharmacological and dietary management <sup>88</sup>.

**Neuroimaging may provide powerful biomarkers.** Neuroimaging has revolutionized neuroscience, facilitating brain-behavior research. Functional magnetic resonance imaging (FMRI) measures brain responses during cognitive-behavioral tasks<sup>89-93</sup>. Arterial spin labeling (ASL) perfusion imaging and magnetic resonance spectroscopy (MRS) enable cerebral blood flow (CBF) and cerebral metabolic dysfunction to be assessed. These MR techniques are noninvasive, have excellent neuroanatomic resolution, and have excellent sensitivity for detecting and measuring subtle functional brain changes over time. Multimodal imaging is being used increasingly clinically, enabling simultaneous measurement of brain structure, function, and pathophysiology. Neuroimaging is relatively inexpensive when performed concurrently and is highly sensitive to treatment effects, <sup>94-102</sup> providing potentially powerful biomarkers for assessing the effects of obesity on brain function and treatment outcomes.

Few neuroimaging studies of weight loss benefits exist. Improved brain health may be possible following weight reduction <sup>16</sup>. Some studies have shown greater white matter integrity <sup>103</sup>, as well as improvements on metabolic indices of oxidative stress and glucose metabolism <sup>75,104</sup> and alterations in FMRI brain response on attention-executive and cue reactivity tasks among people who successfully maintained weight loss <sup>105-107</sup>. A few case reports of neuroimaging show adverse brain effects from bariatric surgery, although these cases are not representative <sup>108-112</sup>. Studies of changes in neuronal function (FMRI), cerebral perfusion (ASL), and metabolic function (MRS) following significant weight loss are needed.

Treatment implications. Findings from this study may lead to new strategies for treating and preventing brain dysfunction, perhaps even slowing the onset of neurodegenerative brain changes <sup>26</sup>. Our findings may eventually influence medical decision-making, particularly if the results suggest that rapid and dramatic weight loss reduces subsequent obesity-related brain dysfunction. The results may also signal a need for additional patient education/training to ensure adherence to postoperative behavioral recommendations. Positive findings would also motivate future research focused on dose-response and whether more modest weight loss via lifestyle intervention or pharmacological treatment produces some benefits for brain health.

**Scientific significance.** The proposed study provides a unique opportunity to examine the effects of severe obesity and surgically induced weight loss on the brain. Past studies of obesity and the brain have largely been either epidemiological or observational. By employing multimodal neuroimaging pre- and post-bariatric surgery, we can

simultaneously assess obesity-associated cerebral metabolite, vascular, and functional disturbances. We will also be able to test the effects of weight loss on brain functions with an approach that can delineate associated cerebral pathophysiology and identify possible mechanisms that cognition improves post-surgery.

We will accomplish several scientific objectives: 1) The study will provide the most comprehensive information to date on the effects of obesity on cerebral metabolic, vascular, and neural functions; 2) The longitudinal design will elucidate the trajectory of cognitive change relative to weight loss and changes in diabetes and metabolite-vascular status; 3) We will determine whether changes in specific risk factors (e.g., diabetes, sleep apnea) mediate these effects; 4) We will explore the potential value of functional neuroimaging indices as biomarkers of subtle cognitive change; 5) We will characterize the relationship between systemic and cerebral inflammatory processes by examining both MRS and serum biomarkers; 6) Bariatric surgery provides a unique experimental approach that goes beyond what can be learned from past observational studies, particularly since significant weight loss will occur relatively quickly and without the intensity of effort required by behavioral interventions; 7) The scientific significance likely extends beyond obesity, providing insights into mechanisms that may contribute to vascular cognitive impairment and cognitive aging, and perhaps even neurodegeneration.

# 5. Specific Aims:

# A. The proposed study is motivated by four broad objectives:

1. To obtain preliminary multimodal *neuroimaging* data on community dwelling adults, including:

<u>Cohort #1</u>- Surgical Candidates for Bariatric Surgery (BMI>35 kg/m<sup>2)</sup> the University of Florida, (goal n=120) with Type 2 Diabetes (60) and Non-Diabetic (60)

<u>Cohort #2</u>- Obese Controls (BMI >35 kg/m<sup>2)</sup> Individuals ages 20+ in the Gainesville community and North Florida region (goal n=60) with Type 2 Diabetes (30) and Non-Diabetic (30) who will not chose Bariatric Surgery

| | Type-2 Diabetes | Non-Diabetic |
|-------------------|-----------------|--------------|
| Bariatric Surgery | N=60 | N=60 |
| Obese Control | N=30 | N=30 |

**Neuroimaging:** The rationale for incorporating neuroimaging is relatively intuitive. There is a compelling need for *in vivo* biomarker discovery and validation for the purposes of *in vivo* biomarkers that can be used to assess brain structure, function and pathophysiology, and that may also be predictive of subsequent functional change as people age, as well as responsive to interventions aimed at preventing cognitive decline, MCI and dementia. There is mounting evidence that vascular and metabolic factors contribute to the development of brain dysfunction in the elderly, and that their effects likely begin long before overt symptoms are apparent. A greater understanding of the influence of these and other risk factors on the aging brain is needed, particularly research directed at underlying neuropathological and potentially modifiable mechanisms linked to these factors. The proposed study will provide preliminary data from several neuroimaging modalities that will

be examined relative physical, social, and cognitive functional measures enabling initial examination of the linkages between these behavioral and physical factors, and cerebral metabolic and hemodynamic function, as well as prodromal structural brain changes in those with and without diabetes, before and after a surgical intervention.

To collect data on the cognitive module of the NIH Toolbox. (See Appendix D for descriptions and summary screen shots)

<u>Cognitive assessment:</u> The rationale for collecting cognitive data using the NIH Tool Box was based on two major considerations:

- 1) NIA has a vested interest in investigators using the Tool Box in large scale studies and randomized controlled trials of the aging brain;
- 2) It was important for purposes of the proposed study to measure cognition at the same time point as the neuroimaging assessment; prior to surgical intervention, 12 weeks post intervention and 18 months post intervention.

This is a new instrument from those currently being employed. The complete cognitive module of the NIH-Toolbox takes approximately 60 minutes and is computerized.

- Dr. Cohen has attended an NIA sponsored meeting in Washington, D.C, in which the Toolbox was unveiled to researchers to determine its psychometric characteristics, feasibility of use and also to reinforce our willingness to consider this for inclusion in this study. Data obtained to date suggests that it is highly reliable and has validity relative to established neuropsychological tests. The assessment approach's inclusion in this large scale study illustrates its relevance in the mission of studying diabetes and metabolic factors affecting health and functional outcomes.
- To collect blood samples from participants for analysis and comparison to other measures previously described.

We will obtain a serum biomarker panel of cytokines and other molecules sensitive to systemic inflammation, metabolic and vascular pathophysiology. Processing will occur in Dr. Leeuwenburgh's laboratory. Potential analyses using Luminex technology include proteonic analysis on cytokines, inflammatory biomarkers, metabolic biomarkers and neurodegenerative biomarkers. Concentrations of the biomarkers will be examined relative to the MRI indices, particularly the proton MRS cerebral metabolites, providing information the correspondence between systemic inflammatory processes evident in the blood and cerebral metabolite disturbances. The MRS indices (choline (Cho), myo-inositol (MI), Nacetyl aspartate (NAA) and glutamate-glutamine (GLX)) provide information regarding neuronal dysfunction and loss and also inflammatory processes occurring in the brain, as described in our previous studies. A blood sample to measure HBA1C (3 month sugar level) will be sent off to Quest Laboratories, with a de-identified participant number only. Because only the CAM-CTRP billing information and a participant number will be submitted, there will be no opportunity for a billing mistake to take place, which protects the participants. 5 mL aliquots of blood will be sent to Avera in South Dakota for genetic sequencing. The data produced by Avera (digital strings of DNA nucleotides), as well as deidentified demographic and comorbidity data from WISE, will be sent to Sarah Medland laboratory in Australia for further analysis. The genetic sequences that result from these analyses are short fragments of DNA from various genes that have relevance to the WISE study (relation to obesity, cognition, etc.). These sequences do not contain enough genetic information to enable for future identification of specific participants. Blood samples and accompanying data will be labeled with only a de-identified participant label and blood will be discarded as biohazardous waste after analysis. As part of our collaboration, the genetic sequences derived by Dr. Sarah Medland in Australia will be entered into a larger database of the ENIGMA obesity workgroup, which contains similar data from investigators around the

- world. This dataset is limited with no PHI, and only a few demographic and clinical diagnostic information.
- 4. To conduct Sleep Apnea Assessments at baseline, to account for obstructive sleep apnea effects on neurocognition, for those who have not been previously assessed and assigned CPAP therapy. The Bariatric Surgery program requires most of its patients to have an overnight in-lab sleep study and CPAP therapy prescribed as needed prior to undergoing surgery. The results of the prescribed sleep study will be obtained from the participant's medical record.
- **B.** The specific study aims are as follows: The goal of the proposed study is to delineate mechanisms underlying the effects of chronic obesity on brain functioning, and the basis for improved neurocognitive performance following bariatric surgery induced weight loss. We will use multimodal neuroimaging methods to determine whether these improvements correspond with enhanced cerebral metabolic or hemodynamic functioning following surgery. We will also examine the contribution of insulin-glucose metabolism, diabetes and sleep apnea to these effects.
  - Aim 1: Demonstrate improved neural function (FMRI) post-surgery compared to obese non-surgical controls. H1: Improved working memory, focused attention and memory recall following bariatric surgery will correspond with increased BOLD response in brain regions of interest (ROIs). On the 2-back working memory paradigm, changes will be greatest in dorsolateral and medial prefrontal cortex (DLPFC and MFC), and the supplementary motor area (SMA). On the CVMT, changes will be greatest in the medial temporal- hippocampal ROIs. H2. Post-surgical changes will persist over 18 months. H3. Baseline cognitive deficits and FMRI abnormalities, greatest among participants with co-morbid diabetes will improve the most, reflecting effects of bariatric surgery on diabetes and metabolic function.
  - Aim 2: Demonstrate that cerebral metabolites (MRS) and perfusion (ASL) improve post-surgically. H1: Cerebral metabolite concentrations will improve in hippocampal and frontal ROIs. Decreased choline (Cho) and Myoinositol (MI) and increased N-acetyl aspartate (NAA) will reflect reduced cerebral inflammation (Cho, MI) and neuronal damage (NAA). H2) Regional cerebral blood flow (ASL) in these same ROIs will increase post-surgically. H3) Cerebral MRS and ASL improvements will be greatest among participants with comorbid diabetes, reflecting benefits of improved glucose metabolism and diabetes status. H4) Cerebral MRS improvements will correspond with reduced concentrations of serum cytokines and other pro-inflammatory/neurotoxic metabolites.
  - Aim 3: Determine whether cerebral metabolite and perfusion effects contribute to enhanced post-surgical cognitive performance and brain function on the FMRI tasks. H1. Cerebral MRS and ASL changes will be shown to mediate enhanced post-surgical neurocognitive and BOLD response. H2. MRS, ASL and FMRI neuroimaging, and serum proinflammatory biomarker improvements at 3 months will be predictive of 18-month change; H3) Post-surgical glucose-insulin changes will also be predictive of improved brain function. H4) While reductions in glucose/insulin disturbances will contribute in part to improved neurocognitive and neural function, weight loss itself, and associated changes in cerebral metabolite and perfusion, will be the strongest predictors of improvements in these functions.
  - **Aim 4:** We will examine the influence of sleep apnea assessed by ambulatory overnight polysomnography (PSG) on obesity-associated brain dysfunction and improvements following weight loss. A sleep apnea severity index will be derived and used as a covariant in the primary analyses for Aims 1-3.

# C. Approach:

Using previously established neuroimaging methods, we will collect *in vivo* MRI measures from participants at the University of Florida McKnight Brain Institute AMRIS facility during a multimodal scanning session in the Phillips 3.0 Tesla scanner, or the UF Health/Shands Siemens 3T MRI Scanner, lasting up to 2 hours, including a short tutorial on the functional task. The primary neuroimaging measures are as follows:

- Structural: cortical and sub-cortical volumes (MPRAGE), white matter hyper-intensity volumes (FLAIR), measure of white matter integrity (DTI)
- MRS: choline (Cho), myo-inositol (MI), N-acetyl aspartate (NAA) and glutamate-glutamine (GLX)) obtained from two primary reagents of interest
- ASL: cerebral blood flow measured from the hippocampus and frontal cortex
- fMRI Active cognitive tasks: continuous visual memory test, working memory test, visual
  matching to sample and others. We will perform FMRI using echo planar BOLD imaging (EPI)
  methods, with data acquired concurrently with ASL

Data from this assessment will provide information regarding brain structural, metabolic/physiological and functional disturbances.

Neurocognitive function will be examined relative to each neuroimaging modality using statistical modeling methods to determine the extent to which they predicts performance in specific cognitive domains (learning-memory, attention-executive, motor-processing speed).

We will also collect a blood sample (approx. 2 TBSP) at the time of the cognitive assessment or MRI visit, which will be stored and analyzed by Dr. Leeuwenburgh's laboratory in the Institute on Aging (IOA) in collaboration with Dr. Cohen to examine how cerebral metabolite abnormalities on MRS (Magnetic Resonance Spectroscopy) correspond with cytokine, ceramide, DNA markers and other metabolic disturbances common to degenerative disease processes.

### 6. Research Plan:

A. Participant Cohorts and Recruitment- We will recruit 200 adult participants (men = 100; women = 100; age: 20-75 years) to obtain and retain an eventual study sample of 180 severely obese adults. The sample will include 120 people from the UF Bariatric Surgery Service undergoing Roux-en-Y Gastric Bypass (RYGB) or gastric sleeve surgery. We will recruit the non-obese controls from the general community. We will recruit both the bariatric surgery and obesity control groups so that approximately 50% of each will have a medical history and current diagnosis of type-2 diabetes based on ADA diagnostic criteria.

| | Type-2 Diabetes | Non-Diabetic |
|-------------------|-----------------|--------------|
| Bariatric Surgery | N=60 | N=60 |
| Obese Control | N=30 | N=30 |

All participants will be informed that the study involves a cognitive assessment, a physical activity questionnaire and assessment, a few cognitive screening measures, the NIH Toolbox of computerized measures, then an MRI session to record images of their brain, and that this will be repeated for a total of 3 study times, Baseline (or Pre-Surgery), 12 weeks, and again between 9 and 18 months Post-Surgery. (See table 1 for details) During the MR session, participants will rest passively in the scanner and also perform approximately 15 minutes of thinking tasks involving attention and memory. They will also be asked to provide a small blood sample (approximately 2 TBSP) for serum biomarkers and blood glucose.

- a. Cohort #1- The surgical candidate group will be presented with the information about the WISE Brain Study, by Recruiting Flyer and if they are interested in participating, will be asked to contact the Program Coordinator, or Recruitment Specialist for more information and screening for the study. In order to undergo bariatric surgery, patients attend an informational bariatric seminar before scheduling a consultation appointment. Patients may be presented information about the study during the seminar but will not be enrolled until after their bariatric consultation appointment. See Appendix NN for the bariatric seminar PowerPoint presentation.
- b. Cohort #2- This group consists of community dwelling obese residents who will not undergo bariatric surgery. Participants will be recruited from the Gainesville area and the North Florida region (target n= 60) by the means of advertisement via IRB approved flyers or by mailing IRB approved letters or postcards and posting on local physical and digital bulletin boards of interest, and newspaper classified ads. Groups may also be recruited by short educational seminars on current research in cognitive aging, with recruitment information made available at the end of the talk. Participants will also be recruited at community events with IRB-approved flyers, and participants will have the option to confidentially provide name, phone number, and email if they wish to be contacted by the study team to determine study eligibility. The contact information will be securely stored during the event and immediately stored in the Cohen Lab per study data safety management plan. In the event that a participant recruited from the bariatric surgery clinic consents to participate but does not have surgery, the participant may be switched to the community cohort.

In addition, participants may be recruited from:

- The Claude D. Pepper Recruitment Registry PI – Dr. Marsiske, IRB # 415-2007
- HealthStreet, IRB # 265-2011
- CAM-CTRP Consent to Contact Registry IRB #133-2013

### B. Inclusion and Exclusion Criteria:

The inclusion criteria for this sample will be aged 20-75yrs. and up, able to walk with or without assistance, with BMI >35, with or without diabetes.

Exclusion of people with pre-existing neurological or psychiatric brain disorders, or MRI exclusions, or diagnosis with a neurodegenerative brain disease like dementia or Alzheimer's or:

- (1) Prior neurological disorder (e.g., dementia, stroke, seizure disorder, traumatic brain injury);
- (2) Montreal Cognitive Assessment (MoCA) score < 17
- For cases in which score is between 17 and 22, Dr. Cohen (PI) will evaluate assessment results and clinical information to make a determination of whether there is evidence of dementia or early neurodegenerative disease. If the data suggests dementia or other neurodegenerative disease, participants will be excluded and referred to the appropriate clinical care.

- (3) Major psychiatric disturbance (e.g., schizophrenia, chronic intractable depression, substance abuse);
- (4) Severe CVD history based on criteria described below (e.g. coronary heart disease, coronary revascularization procedure, peripheral vascular disease);
- (5) Unstable medical conditions (e.g. cancer; basal cell skin and limited prostate cancer are acceptable);
- (6) MRI contraindications (e.g., pregnancy, claustrophobia, metal implants, circumference > 60 cm, weight > 550 lbs); Additional criteria involve being eligible for a MRI scan; People who have metal implants, who are claustrophobic, or do not meet other standard MR safety screening criteria per screening form (Appendix A) will not be included in the MRI portion of the study.
- (7) Females of child-bearing potential (younger than 62 years old and no previous hysterectomy) will be screened for pregnancy prior to each MRI session (using urine hCG pregnancy test) and women whose test results read as "positive" will be excluded from study participation.
- (8) Physical impairment precluding motor response or lying still on back for 1 hr.

Participants who cannot participate in the MRI due to weight/size limitations will be temporarily excluded from that portion of the study and will be asked to complete only the cognitive assessments, physical tasks, and blood draw at the baseline visit. These participants will be reassessed for MRI eligibility at the 12-week follow-up visit. No MRI data will be collected from participants who exceed weight/size limitations after the 12 week follow up.

C. Safety monitoring: All participants will be screened for MRI safety prior to undergoing MR imaging, or entering the MR suite. The subject safety screening documents utilized at the University of Florida Advanced Magnetic Resonance Imaging and Spectroscopy (AMRIS) facility and UFHealth/Shands are attached as Appendix A to this proposal, and will be used as a screening tool for the study.

### D. Referrals:

- a. MRI findings: If any questionable findings are noted on the MRI scan by the study team, the study's PI will be notified. The study team and/or PI will contact participants to notify them of the incidental findings, provide them with copy of their MRI scan and will encourage follow-up with their primary care physician.
- b. Mental Health Issues: If any assessments or conversations with participants indicate depression, or other new mental health or cognitive functioning concerns, they will be immediately reported to the PI, and the PI will phone the participant to offer referral for appropriate clinical care.
- **c. Post-Surgical complaints:** Should participant discuss any post-surgical adverse events that are related to the surgery, the PI will be notified, and call the participant to encourage follow-up with their clinician, surgeon, or internist, or referrals made as needed.
- d. **Sleep Disorders:** If any sleep disorders are discovered by the sleep study research team, the Sleep Disorder Referral Letter will be sent to the participant. This will strongly encourage the participant to seek additional medical treatment, but will not exclude them from future participation in the study. See Appendices on Sleep Documents section AA.
- **E.** Participant Copy of MR Scan- After the long-term follow-up MRI scan, we will provide a copy of the MR scan for participants to keep as a courtesy for their records. Participants are informed on the Informed Consent Form that this scan is not for diagnostic purposes, but for research analysis only, and that no "results" will be made available with the scan. Participants are encouraged to share the scan with their physician to keep on file for their records only.

### F. Procedural Sequence for Study Visit:

# **Study Overview**

Occurs at baseline, 12 weeks and 9 to 18 months

#### Recruitment and Screening (baseline only)

Recruitment Processes PreScreen Informed Consent Inclusion/Exclusion Screen

#### **Assessment**

Demographic Information
Medical/Psychosocial history
Neurocognitive Assessments
Psychiatric/Behavioral Measures
Pain Questionnaire
Sleep Questionnaire
Weight loss questionnaire
Blood Draw for Biomarkers and Glucose
Optional Stool Sample

#### MR Assessment

Anatomical and Functional Brain Scan

- a. Potential participants will be pre-screened at the time of their initial contact for information about the study, either over the phone or in a private location Participants may also be contacted by email to set up a phone screening. (See Appendix K- Telephone Pre-Screen and Appendix JJ.2 Email to Interested Candidates).
- b. Potential participants identified in person will be asked to complete the WISE Brain Study Screening Informed Consent in order to begin their participation. This ICF will allow study staff to determine eligibility for the study and schedule study-related visits in coordination with the participants' clinical care. Participants who screen in will be invited back to complete the full ICF and complete the remainder of the study activities.
- c. If participant meets all inclusionary guidelines, they will be scheduled for their preferred study visit appointments in coordination with their surgery (if applicable).
- d. Participants will be explained the study activities again, and the Full Informed Consent will be reviewed with them in a private location. Participants will have as much time as needed to discuss the information with their friends and family. They will be given time to consider enrollment in the study. They will have many opportunities to ask questions and get those questions answered prior to giving their official consent to participate.
- e. After informed consent is documented, participants will be screened for inclusion/exclusion factors, including pregnancy.
- f. Participants may have the MRI Measurement Device (See Appendix AA.2 in Misc. Attachments) demonstrated for them to visually see the size of the inside of the chamber of the MRI Scanner. Participants may be asked to try the device on themselves to gain a greater understanding of the size constraints related to the MRI Scan, and to give them a chance to experience the snug fit inside the core of the scanner. If participants can not fit in the measurement device, they will be thanked for their limited participation, and given a \$10 pre-paid debit card to thank them for their time and effort.
- g. Participants will be given a Medical History evaluation, using the Medical History Form. (See Appendix C)
- h. Participants will be assessed on cognitive ability, using the MoCA, CVLT-2, PASAT and Boston naming, commonly used in the assessment of MCI and early dementia, and included on the IRB list of approved Psychological Measures. They will also be administered the NIH Toolbox Cognitive performance measures listed in Table 1 (See Appendix D for samples) This portion will take approximately 3 1/2 hours and thus a portion may be done at the time for their MRI visit.

- i. We would like to audio record the cognitive sessions for quality assurance. These recordings are for the examiners to accurately note participant's responses and score assessments. The audio recordings will be securely storage in our study's secure computer system. Only research assistants and coordinators who have conducted the study visit will have access to them. The recordings will be deleted upon their attended use.
- a. A research study staff certified phlebotomist will obtain the blood sample. Approximately (2TBSP. or less) of blood will be obtained from each participant and stored for analysis of metabolic biomarker panels, inflammatory and neurodegenerative biomarkers and cytokines, along with genomic analysis. Some of the blood specimens could be sent to study collaborators for further analysis. These samples will be coded and will not have any PHI associated with them. These collaborators will have signed Confidentiality Agreements with UF to secure privacy. You will not get any information back regarding these blood tests; they are only being done for the purposes of this research. De-identified blood samples will be sent to Avera in North Dakota for genetic sequencing. Resulting data, along with deidentified demographic and comorbidity data, will then be sent to Sarah Medland laboratory in Australia, where analyses will be conducted on the genetic sequences to reduce the data to DNA coding of genes that have previously been shown to be of relevance to obesity and cognition. Data and samples will only be labelled with the participant's study ID and blood will be discarded as biohazardous waste after analysis. Genetic sequences derived by Dr. Sarah Medland in Australia will be entered into a larger database of the ENIGMA obesity workgroup. Only de-identified data and sparse demographic and clinical information is entered into the database. We will also look at the sugar levels you have in your blood as a result of your body's processing the food that you eat. Blood specimens will be sent to Quest Diagnostics for this test. The specimens will be coded.
- b. Participants may be asked to provide an optional stool sample at baseline, 12-week, and 9 to 18-month follow-up visits. The stool sample may be provided by the participant at any time during the study visit or may be collected at home. If the sample is not returned within 48 hours of its collection, study staff will contact the participant to remind them to return the sample. The sample will be collected using a kit that fits over a toilet, and includes a sterile spatula in which the participant will obtain an approximately 50cc scoop of their stool and place in container included in the collection kit. A biohazard specimen transport bag and a brown paper bag will be provided to ensure proper transport and discretion. Included in the collection kit is the Bristol Stool Chart where participants can identify the type of stool produced during collection.
- c. A take home packet of questionnaires may be sent home with participant, to save them time at the study visit. This packet can be returned at their next visit. The take home packet can include items such as:
  - i. Medication List
  - ii. Baecke- activity survey
  - iii. Beck Depression Inventory (BDI-II)
  - iv. Charlson Comorbidity survey
  - v. CHAMPS- physical activity survey
  - vi. Epworth Sleepiness Scale
  - vii. SF-36 Lifestyle Activity
  - viii. TFEQ Eating Inventory
  - ix. Pain Questionnaire
  - x. Weight loss questionnaire
  - xi. UCLA Loneliness questionnaire
  - xii. Trait Anxiety Inventory for Adults (STAI)
  - xiii. Eating Disorders Inventory-2 (EDI-2)
  - xiv. Binge Eating Scale
  - xv. Marlowe-Crowne Social Desirability Scale
  - xvi. Master Questionnaire- Revised

The following procedures will take place at the AMRIS Center at the McKnight Brain Institute or the UFHealth Shands Siemens 3T scanner - and can be completed at a separate visit if preferred.

d. Participants will be accompanied by study staff to the UFHealth Shands Siemens 3T Scanner which has a larger bore size, (for larger sized participants) where neuroimaging will be performed for approximately one hour. During the scanning session, brain MRI and MRS data will be obtained using a series of sequences in a pre-constructed imaging protocol: 1) T1 MPRAGE; 2) FLAIR; 3) DTI; 4) MRS-Frontal Voxel; 5) MRS-Hippocampal voxel; 6) ASL; 7) Resting BOLD. ASL and BOLD sequences will be interleaved to reduce the required time.

### Participant Retention Plan:

In an effort to maximize study retention, letters and thank you-notes may be sent to a participant's home during follow-up periods or if a participant cannot be reached by telephone to schedule his/her next visit. Participants will be mailed or emailed visit confirmations with directions. See Appendix JJ.

We may also contact participants by phone in order to ask general questions about well-being and ability to continue participation in order to maintain contact during follow-up periods. See Appendix KK.

A newsletter discussing study progress and other potential items of interest to the study population will be mailed quarterly to all enrolled participants. See Appendix LL.

We will offer items stamped with the study logo that may support the participants in their daily lives, particularly post-bariatric surgery, at specific time points throughout the study. See Appendix MM for gift schedule.

### G. Compensation:

### Screen Fail:

If a participant arrives for an appointment, but does not pass the screening measures for the MoCA (score < 20) or the MRI (pregnancy, size, or claustrophobia), they will be given a \$10 pre-paid debit card to thank them for their limited participation.

**Participation in study activity:** Participants that complete the cognitive assessment portion of the visit will be given a \$60 pre-paid debit card to compensate them for their time and effort. If they participate in the blood draw, they will also receive a \$15 pre-paid debit card to compensate them for time and effort. If they participate in the optional stool sample, they will receive a \$15 pre-paid debit card to compensate them for time and effort. Finally, participants that complete the MR portion of the visit will be given a pre-paid debit card for \$60 for each scan to compensate them for time and effort. This compensation system will be the same for all 3 times that the participant comes to participate in research, Baseline, 12 weeks Post surgery, and at 9 to 18 months Post Surgery.

**Travel:** If they have traveled 20 miles or more (one way), they will receive an additional \$10 prepaid debit card at each visit to compensate them for additional gas expense.

- **H.** *Data Storage:* There are 5 areas of data collection which will be stored. All data will be coded to protect the PHI of participants. That coded information will be kept in a secure area, with a locked door.
  - MRI scans/images- These images will be stored on password protected computers and encrypted 4T storage drives. Any DVD disks or memory sticks with image data will be coded, locked in a secure room, and in a locked area. This data will also be stored on secure UF servers associated with the UF HiPerGator system, with all PHI removed.

- 2. NIH Toolbox Results- This web based program transmits the study identifier coded data directly back to the NIH Toolbox servers, and is not stored locally. The PHI free, coded data is then returned to UF and stored on password protected, encrypted computers.
- 3. Cognitive Assessments done locally- This data will be coded by study participant number, and kept in a secure location in a locked room. Data may be entered into a Redcap Database system or similar database system for analysis.
- 4. Blood- The blood will be coded, PHI removed, and be stored in a secure lab area, overseen by Dr. Leeuwenburgh.
- 5. Stool- All stool samples will be de-identified and labeled only with the WISE Study ID# before transfer to the analyses site. There is not a way for offsite collaborators to link the samples to the participants. Research staff will then place a preprinted label on the stool collection vial with the study ID#.

# 7. Possible Discomforts and Risks

**Participant Burden**: Participants will experience at least two study visits at each time point, BL, 12 weeks, and 9 to 18 months, depending on their choice and availability. It will consist of a few cognitive measures, a physical activity questionnaire, approximately 1.5 hour cognitive assessment that includes the NIH Toolbox Cognitive measures, 20 minute physical activity measures, one or two one hour MR imaging sessions with two thinking tasks, and a blood draw. During the MR scanning, several sequences will be obtained while participants passively rest in the scanner. Active fMRI tasks will also be administered though this will be limited to approximately 15 minutes. They may also be asked to fill out questionnaires at home and bring them to their next visit.

**MRI:** During the MRI procedure, participants will be able to talk with the MRI staff through a radio intercom speaker system, and, in the event of an emergency, they can tell them to stop the scan immediately. Participants will be asked frequently during the preparation and scanning period whether they are experiencing any discomfort, and corrections will be made as necessary.

Participants may experience discomfort during the scanning process due to limited space inside the bore of the magnet. Subjects will be closely monitored and repeatedly checked by the investigators to ensure comfort. Participants may also become uncomfortable from lying still for an extended period of time, or if they do not like to be in close spaces (have "claustrophobia"). Padding with blankets can be used to prevent discomfort while lying in the magnet.

The MRI scanner produces a loud "hammering" noise, which has been reported to produce temporary hearing loss in a very small number of people. Participants will be provided with earplugs to wear in the scanner, and also headphones to reduce this risk and possible discomfort.

**Blood Draw:** The risks of drawing blood from a vein include discomfort at the site of puncture; possible bruising and swelling around the puncture site; rarely an infection; and, uncommonly, faintness from the procedure. These risks will be minimized by utilizing only trained personnel for drawing blood and using sterile and disposable materials.

**Stool Sample:** The process of collecting a stool specimen, while potentially messy, has no risk beyond normal bathroom activity. Participants will be provided with the stool collection kit and protective material (gloves, etc) at no cost to them. Our research team will provide instructions regarding the process. Persons can either bring the sample form home, or they can provide it during the day of their study visits (using a bathroom at the research facilities). A demonstration kit will be available during the study visit to show the components and staff will also instruct participants on how to properly seal the bio bag to prevent contamination during transportation. Participants may elect to collect the sample at home to reduce embarrassment.

**Computer based tests:** There is a risk that participants will find memory and concentration tests to be difficult, or frustrating, because it is a new task that they are not familiar with, and may be challenging to

their thinking and memory. Participants may skip any question they do not wish to answer. Research staff will explain what to do and help them do the tasks during their research visit.

**PHI:** Researchers will take appropriate steps to protect any information they collect about study participants. However, there is a slight risk that information about them could be revealed inappropriately or accidentally. Depending on the nature of the information, such a release could upset or embarrass participants, or possibly affect their insurability or employability. These risks will be minimized by storing study documents in secure locations and electronic files on servers protected by passwords; only authorized personnel will have access to the study documents and files.

**COVID-19:** Upon arriving at the lab space, researchers will use one of several touchless thermometers to take their temperature. If their temperature is 100.4 degrees Fahrenheit or greater, they will leave immediately and inform the PI. Researchers are required to wear surgical masks and gloves, both of which are available within the lab space. Before beginning a participant visit, researchers will use soap and water to clean any frequently used surfaces, such as door handles and tables. These surfaces will then be sanitized with Clorox wipes; items that can't first be cleaned with soap and water, such as electronics, will only be wiped down with Clorox wipes.

Researchers will greet participants outside the building and ask a series of screening questions to determine if the participant currently has any symptoms indicative of COVID-19, has recently traveled to an area with known local spread of COVID-19, or has come into close contact with someone with a laboratory-confirmed COVID-19 diagnosis. If the answer is yes to any of these questions, the participant will not be allowed to complete their visit until they are tested for the virus. If the participant did travel to a known area of COVID-19, but it was more than 14 days prior to participant examination and the participant is symptom free, the examination will be allowed. Researchers will also measure the participant's temperature using the touchless thermometer. If the participants' temperature is 100.4 degrees Fahrenheit or greater, the examination will not be allowed.

If participants arrive without a surgical mask and gloves, the researcher will provide them with both before entering the building. Researchers and participants will remain 6 feet apart throughout the visit, using red tape marks on the floor to indicate where each person should sit. If either the researcher or participant needs to drink, they will step outside and away from people to remove their mask and drink. If the participant needs to use the restroom, they will be asked to remove their gloves and use new gloves when they return. After the visit, the researcher will again clean the testing room with Clorox wipes, making sure to disinfect any surfaces that they or the participant may have touched. Gloves will be discarded in biohazard bins.

Participants and study staff are required to wear a mask at the UF Health Shands MRI Suite. Researchers will maintain a 6-foot distance between themselves and participants at all times. Study materials, including laptop, laptop bag, joystick for task, etc., will be cleaned with Clorox wipes before and after each participant. Masks will also be required within the MRI scanner; the hospital will provide masks that do not contain metal for participant safety.

# 8. Possible Benefits:

There are no direct benefits to subjects from participating in this study. Results from this study may benefit future researchers and physicians with the diagnosis and prevention of cognitive decline and other brain pathologies related to diabetes.

# 9. Conflicts of Interest:

There are no conflicts of interest.

# **Tables and Appendices:**

### Table 1- Cognitive Measures and Surveys

Appendix A- AMRIS and UFHealth Shands MRI Procedure Screening Form for study participants

- B- WISE Brain Study Inclusion/Exclusion
- C- Medical History Questionnaire
- D- NIH Toolbox Screenshots & Description
- E- Physical Activity Questionnaire CHAMPS
- F- N-back and CVMT task samples
- G- Parking directions
- K- Telephone Pre-Screening Script
- N- MoCA
- O-COWA
- P- Physical Measures Six Minute Walking and SPPB
- Q- Eating Inventory (TFEQ)
- R- Baecke Physical Activity Questionnaire
- S- Pain Questionnaire
- T- Medical Outcomes, SF-36
- U- Medication list
- V- Weight Loss Questionnaire
- W- Epworth Sleep Scale
- X- MRI Appointment Information Form
- Y- WISE Homework Letter
- Z- Sleep Lab Documents
  - Z.1 Sleep Lab Map
  - Z.2 Sleep Lab Directions
  - Z.3 Sleep Disorder Referral Form
  - Z.4 PSG instructions
  - Z.5 PSG Pre-visit instructions
  - Z.6 PSG Return Agreement

### AA- MRI Documents

- AA.1 Participant Information
- AA.2 MRI Measurement Tool
- AA.3 MRI Mock Scanner
- BB- Pre-Paid Debit Card Payment Form
- CC- Adaptive Rate Continuous Performance Task
- DD- UCLA Loneliness Scale
- EE- Trait Anxiety Inventory for Adults (STAI)
- FF Eating Disorders Inventory-2 (EDI-2)
- GG Binge Eating Scale
- HH Marlowe-Crowne Social Desirability Scale
- II Master Questionnaire- Revised
- JJ Participant Communication Materials
  - JJ.1 Thank you card
  - JJ.2 Email for Interested Candidates
  - JJ.3 WISE Brain Study Timeline Community Participant
  - JJ.4 WISE Brain Study Timeline Surgical Participant
  - JJ.5 Letter to be Mailed between Visits 2 and 3
  - JJ.6 Letter for Difficult to Contact Participants
  - JJ.7 Final Letter for Difficult to Contact Participants
  - JJ.8 Reminder card
  - JJ.9 Letter/Email for Visit Confirmations at CRC
  - JJ.10 Letter/Email for Visit Confirmations at MBI

# JJ.11 Parking and Directions to CRC JJ. 12 Directions to UF McKnight Brain Institute

KK – WISE Follow Up Phone Questionnaire

LL – WISE Spring 2017 Newsletter MM – Gift Schedule and Items

NN - Bariatric Seminar Presentation

| Table 1. Activity Summary including Cognitive Measures and Surveys | | Cohort<br>#1<br>Surgical<br>Candidates | Cohort<br>#2<br>NonSurgical<br>Candidates |
|---|---|---|---|
| Telephone Pre Screen | Appendix K | ✓ | ✓ |
| Part #1 of Study Visit: | | | |
| Pre-Scan Screening & | | | |
| Assessments | | | |
| MoCA | Appendix N | ✓ | ✓ |
| COWA | Appendix O | ✓ | ✓ |
| MRI Screening | Appendix A | ✓ | ✓ |
| Pregnancy Test | If required - female <62 | ✓ | ✓ |
| Medical Health History | Appendix C | ✓ | ✓ |
| Medication list | Appendix U | ✓ | ✓ |
| Medical Outcomes SF-36 | Appendix T | ✓ | ✓ |
| Physical Activity Questionnaire (CHAMPS) | Appendix E | <b>✓</b> | <b>✓</b> |
| Boston Naming Test | Approved IRB Psych list | ✓ | ✓ |
| CVLT | Approved IRB Psych List | ✓ | ✓ |
| Beck Depression Inventory | Approved IRB Psych List | ✓ | ✓ |
| Stroop | Approved IRB Psych List | ✓ | ✓ |
| Trails | Approved IRB Psych List | ✓ | ✓ |
| Adaptive Continuous | Appendix DD | ✓ | ✓ |
| Performance Task | PP | | |
| Paced Auditory Serial Addition | Approved IRB Psych list | ✓ | ✓ |
| Test | | | |
| Eating Inventory (TFEQ) | Appendix Q | ✓ | ✓ |
| Baecke Questionnaire | Appendix R | ✓ | ✓ |
| Weight Loss Questionnaire | Appendix V | ✓ | ✓ |
| Home Polysomnography | Provided by UF Sleep Study Lab | ✓ | ✓ |
| Assessment Instructions | | | |
| Epworth Sleep Scale | Appendix W | ✓ | ✓ |
| Physical Measures (6MW, SPPB) | Appendix P | <b>✓</b> | <b>√</b> |
| Pain Questionnaire | Appendix S | ✓ | ✓ |
| UCLA Loneliness | Appendix DD | <b>√</b> | ✓ |
| Trait Anxiety Inventory for Adults | Appendix EE | <b>√</b> | <b>√</b> |
| (STAI) | | | |
| Eating Disorders Inventory-2 (EDI-2) | Appendix FF | ~ | ✓ |
| Binge Eating Scale | Appendix GG | ✓ | ✓ |
| Marlowe-Crowne Social | Appendix HH | ✓ | <b>√</b> |
| Desirability Scale | | | |
| Master Questionnaire- Revised | Appendix II | ✓ | ✓ |
| Blood Draw | | | |
| Blood Serum for Biomarkers | | ✓ | ✓ |

| All NIH Toolbox Samples: | See Appendix D | | |
|---|---|---|---|
| Dimensional Change Card Sort | NIH Tool Box – Executive | ✓ | ✓ |
| Flanker | NIH Tool Box – Attention/Executive | ✓ | ✓ |
| Picture Sequence | NIH Tool Box – Working Memory | ✓ | ✓ |
| Auditory Verbal Learning (Rey) | NIH Tool Box – Episodic Memory | ✓ | ✓ |
| Picture Vocabulary | NIH Tool Box – Language | ✓ | ✓ |
| Oral Reading Recognition | NIH Tool Box - Language | ✓ | ✓ |
| Pattern Comparison | NIH Tool Box- Processing Speed | ✓ | ✓ |
| Oral Symbol Digit | NIH Tool Box- Processing Speed | ✓ | ✓ |
| List Sorting | NIH Tool Box- Working Memory | ✓ | ✓ |
| Part #2 of Study Visit: | | | |
| Pregnancy Test | If required - female <62 | ✓ | ✓ |
| MRI Brain Scan | | ✓ | ✓ |
| Functional Tasks in MRI | | | |
| Continuous Visual Learning | See Appendix F | ✓ | <b>√</b> |
| Memory CVMT | | | |
| N-Back Measure | See Appendix F | <b>√</b> | <b>√</b> |

### **Literature Cited:**

- 1. Main ML, Rao SC, O'Keefe JH. Trends in obesity and extreme obesity among US adults. JAMA 2010;303:1695; author reply -6.
- 2. Ogden CL, Carroll MD, Curtin LR, McDowell MA, Tabak CJ, Flegal KM. Prevalence of overweight and obesity in the United States, 1999-2004. JAMA 2006;295:1549-55.
- 3. Vastag B. Obesity Is Now on Everyone's Plate. JAMA 2004;291:1186-8.
- 4. Manson JE, Bassuk SS. Obesity in the United States: a fresh look at its high toll. JAMA 2003;289:229-30.
- 5. Hebert L, Scherr PA, Bienias JL, Bennett DA, Evans DA. Archives of Neurology. Alzheimer disease in the US population: prevalence estimates using the 2000 census. Arch Neurol 2003;60::1119-22.
- 6. 2009 Alzheimer's disease facts and figures. Alzheimers Dement 2009;5:234-70.
- 7. Kalmijn S, Foley D, White L, et al. Metabolic cardiovascular syndrome and risk of dementia in Japanese-American elderly men. The Honolulu-Asia aging study. Arterioscler Thromb Vasc Biol 2000;20:2255-60.
- 8. De Leeuw FE, Barkhof F, Scheltens P. Alzheimer's disease--one clinical syndrome, two radiological expressions: a study on blood pressure. J Neurol Neurosurg Psychiatry 2004;75:1270-4.
- 9. Majeski EI, Widener CE, Basile J. Hypertension and dementia: does blood pressure control favorably affect cognition? Curr Hypertens Rep 2004;6:357-62.
- 10. Petersen RC, Smith GE, Waring SC, Ivnik RJ, Tangalos EG, Kokmen E. Mild cognitive impairment: clinical characterization and outcome. Arch Neurol 1999;56:303-8.
- 11. Tervo S, Kivipelto M, Hanninen T, et al. Incidence and risk factors for mild cognitive impairment: a population-based three-year follow-up study of cognitively healthy elderly subjects. Dement Geriatr Cogn Disord 2004;17:196-203.
- 12. Breteler MM. Vascular risk factors for Alzheimer's disease: an epidemiologic perspective. Neurobiol Aging 2000;21:153-60.
- 13. Luchsinger JA, Reitz C, Honig LS, Tang MX, Shea S, Mayeux R. Aggregation of vascular risk factors and risk of incident Alzheimer disease. Neurology 2005;65:545-51.
- 14. Riekse RG, Leverenz JB, McCormick W, et al. Effect of vascular lesions on cognition in Alzheimer's disease: a community-based study. J Am Geriatr Soc 2004;52:1442-8.
- 15. Bhargava D, Weiner MF, Hynan LS, Diaz-Arrastia R, Lipton AM. Vascular disease and risk factors, rate of progression, and survival in Alzheimer's disease. J Geriatr Psychiatry Neurol 2006;19:78-82.

- 16. Gunstad J, Strain G, Devlin MJ, Wing R, Cohen RA, Paul RH, Crosby RD, Mitchell JE. Improved Memory Function 12 Weeks after Bariatric Surgery. Surgery for Obesity and Related Diseases In press.
- 17. Miller LA, Crosby RD, Galioto R, et al. Bariatric Surgery Patients Exhibit Improved Memory Function 12 Months Postoperatively. Obes Surg 2013.
- 18. Alosco ML, Spitznagel MB, Strain G, et al. Improved memory function two years after bariatric surgery. Obesity (Silver Spring) 2013.
- 19. Cohen RA, Poppas A, Forman DE, et al. Vascular and cognitive functions associated with cardiovascular disease in the elderly. J Clin Exp Neuropsychol 2009;31:96-110.
- 20. Gunstad J, Cohen RA, Tate DF, et al. Blood pressure variability and white matter hyperintensities in older adults with cardiovascular disease. Blood Press 2005;14:353-8.
- 21. Hoth K, Tate DF, Poppas, A, Forman DE, Gunstad J, Moser DJ, Paul RH, Jefferson AL, Haley AP, Cohen RA. Endothelial function and whiter matter hyperintensities in older patients with cardiovascular disease. Stroke In Press.
- 22. Jefferson AL, Holland CM, Tate DF, et al. Atlas-derived perfusion correlates of white matter hyperintensities in patients with reduced cardiac output. Neurobiol Aging 2009.
- 23. Jefferson AL, Tate DF, Poppas A, et al. Lower cardiac output is associated with greater white matter hyperintensities in older adults with cardiovascular disease. J Am Geriatr Soc 2007;55:1044-8.
- 24. Paul RH, Gunstad J, Poppas A, et al. Neuroimaging and cardiac correlates of cognitive function among patients with cardiac disease. Cerebrovasc Dis 2005;20:129-33.
- 25. Morris JC, Storandt M, Miller JP, et al. Mild cognitive impairment represents early-stage Alzheimer disease. Arch Neurol 2001;58:397-405.
- 26. Cardiovascular disease statistics American Heart Association 2004. (Accessed at
- 27. Prevalence of obesity among adults with arthritis --- United States, 2003--2009. MMWR Morb Mortal Wkly Rep 2011;60:509-13.
- 28. Curtis LH, Hammill BG, Bethel MA, Anstrom KJ, Gottdiener JS, Schulman KA. Costs of the metabolic syndrome in elderly individuals: findings from the Cardiovascular Health Study. Diabetes care 2007;30:2553-8.
- 29. Barkin SL, Heerman WJ, Warren MD, Rennhoff C. Millennials and the World of Work: The Impact of Obesity on Health and Productivity. Journal of business and psychology;25:239-45.
- 30. Kushner RF, Foster GD. Obesity and quality of life. Nutrition 2000;16:947-52.
- 31. Bose K. Age trends in adiposity and central body fat distribution among adult white men resident in Peterborough, East Anglia, England. Collegium antropologicum 2002;26:179-86.
- 32. Houston DK, Ding J, Nicklas BJ, et al. The association between weight history and physical performance in the Health, Aging and Body Composition study. International journal of obesity (2005) 2007;31:1680-7.
- 33. Wyatt SB, Winters KP, Dubbert PM. Overweight and obesity: prevalence, consequences, and causes of a growing public health problem. The American journal of the medical sciences 2006;331:166-74.
- 34. Prevalence of overweight and obesity among adults with diagnosed diabetes--United States, 1988-1994 and 1999-2002. MMWR Morb Mortal Wkly Rep 2004;53:1066-8.
- 35. Prevalence of chronic kidney disease and associated risk factors--United States, 1999-2004. MMWR Morb Mortal Wkly Rep 2007;56:161-5.
- 36. State-specific incidence of diabetes among adults--participating states, 1995-1997 and 2005-2007. MMWR Morb Mortal Wkly Rep 2008;57:1169-73.
- 37. Differences in prevalence of obesity among black, white, and Hispanic adults United States, 2006-2008. MMWR Morb Mortal Wkly Rep 2009;58:740-4.
- 38. Prevalence of abnormal lipid levels among youths --- United States, 1999-2006. MMWR Morb Mortal Wkly Rep 2010;59:29-33.
- 39. Daviglus ML, Talavera GA, Aviles-Santa ML, et al. Prevalence of major cardiovascular risk factors and cardiovascular diseases among Hispanic/Latino individuals of diverse backgrounds in the United States. JAMA 2012;308:1775-84.
- 40. Wijeysundera HC, Machado M, Farahati F, et al. Association of temporal trends in risk factors and treatment uptake with coronary heart disease mortality, 1994-2005. JAMA 2010;303:1841-7.

- 41. McTigue K, Larson JC, Valoski A, et al. Mortality and cardiac and vascular outcomes in extremely obese women. JAMA 2006;296:79-86.
- 42. Cohen RA, Moser DJ, Clark MM, et al. Neurocognitive functioning and improvement in quality of life following participation in cardiac rehabilitation. Am J Cardiol 1999;83:1374-8.
- 43. Osowiecki DM, Cohen RA, Morrow KM, et al. Neurocognitive and psychological contributions to quality of life in HIV-1-infected women. AIDS (London, England) 2000;14:1327-32.
- 44. Al-Khindi T, Macdonald RL, Schweizer TA. Cognitive and functional outcome after aneurysmal subarachnoid hemorrhage. Stroke;41:e519-36.
- 45. Wadley VG, Crowe M, Marsiske M, et al. Changes in everyday function in individuals with psychometrically defined mild cognitive impairment in the Advanced Cognitive Training for Independent and Vital Elderly Study. J Am Geriatr Soc 2007;55:1192-8.
- 46. Soderqvist A, Miedel R, Ponzer S, Tidermark J. The influence of cognitive function on outcome after a hip fracture. The Journal of bone and joint surgery 2006;88:2115-23.
- 47. Brook JS, Zhang C, Saar NS, Brook DW. Psychosocial predictors, higher body mass index, and aspects of neurocognitive dysfunction. Perceptual and motor skills 2009;108:181-95.
- 48. Ettenhofer ML, Hinkin CH, Castellon SA, et al. Aging, neurocognition, and medication adherence in HIV infection. Am J Geriatr Psychiatry 2009;17:281-90.
- 49. Ochner CN, Green D, van Steenburgh JJ, Kounios J, Lowe MR. Asymmetric prefrontal cortex activation in relation to markers of overeating in obese humans. Appetite 2009;53:44-9.
- 50. Yerramasu A, Dey D, Venuraju S, et al. Increased volume of epicardial fat is an independent risk factor for accelerated progression of sub-clinical coronary atherosclerosis. Atherosclerosis 2012;220:223-30.
- 51. Irzmanski R, Sliwczynska-Rodziewicz D, Pawlicki L, Kowalski J. The influence of risk factors for metabolic syndrome on vascular complications. Angiology 2012;63:86-91.
- 52. Wildman RP, Kaplan R, Manson JE, et al. Body size phenotypes and inflammation in the Women's Health Initiative Observational Study. Obesity (Silver Spring) 2011;19:1482-91.
- 53. Liu H, Zhang X, Feng X, Li J, Hu M, Yambe T. Effects of metabolic syndrome on cardio-ankle vascular index in middle-aged and elderly Chinese. Metab Syndr Relat Disord 2011;9:105-10.
- 54. Leiter LA, Fitchett DH, Gilbert RE, et al. Cardiometabolic risk in Canada: a detailed analysis and position paper by the cardiometabolic risk working group. Can J Cardiol 2011;27:e1-e33.
- 55. Wild RA, Carmina E, Diamanti-Kandarakis E, et al. Assessment of cardiovascular risk and prevention of cardiovascular disease in women with the polycystic ovary syndrome: a consensus statement by the Androgen Excess and Polycystic Ovary Syndrome (AE-PCOS) Society. J Clin Endocrinol Metab 2010;95:2038-49.
- 56. Solomon A, Christian BF, Norton GR, Woodiwiss AJ, Dessein PH. Risk factor profiles for atherosclerotic cardiovascular disease in black and other Africans with established rheumatoid arthritis. J Rheumatol 2010;37:953-60.
- 57. Sakurai T, Iimuro S, Araki A, et al. Age-associated increase in abdominal obesity and insulin resistance, and usefulness of AHA/NHLBI definition of metabolic syndrome for predicting cardiovascular disease in Japanese elderly with type 2 diabetes mellitus. Gerontology 2010;56:141-9.
- 58. Frisardi V, Solfrizzi V, Seripa D, et al. Metabolic-cognitive syndrome: a cross-talk between metabolic syndrome and Alzheimer's disease. Ageing Res Rev 2010;9:399-417.
- 59. Maher PA, Schubert DR. Metabolic links between diabetes and Alzheimer's disease. Expert Rev Neurother 2009;9:617-30.
- 60. Craft S. The role of metabolic disorders in Alzheimer disease and vascular dementia: two roads converged. Arch Neurol 2009;66:300-5.
- 61. Gunstad J, Keary TA, Spitznagel MB, et al. Blood pressure and cognitive function in older adults with cardiovascular disease. Int J Neurosci 2009;119:2228-42.
- 62. Tate DF, Jefferson AL, Brickman AM, et al. Regional White Matter Signal Abnormalities and Cognitive Correlates Among Geriatric Patients with Treated Cardiovascular Disease. Brain Imaging Behav 2008;2:200-6.
- 63. Gunstad J, Benitez A, Hoth KF, et al. P-selectin 1087G/A polymorphism is associated with neuropsychological test performance in older adults with cardiovascular disease. Stroke 2009;40:2969-72.

- 64. Hoth KF, Tate DF, Poppas A, et al. Endothelial function and white matter hyperintensities in older adults with cardiovascular disease. Stroke 2007;38:308-12.
- 65. Haley AP, Forman DE, Poppas A, et al. Carotid artery intima-media thickness and cognition in cardiovascular disease. Int J Cardiol 2007;121:148-54.
- 66. Gunstad J, Schofield P, Paul RH, et al. BDNF Val66Met polymorphism is associated with body mass index in healthy adults. Neuropsychobiology 2006;53:153-6.
- 67. Paul RH, Haque O, Gunstad J, et al. Subcortical hyperintensities impact cognitive function among a select subset of healthy elderly. Arch Clin Neuropsychol 2005;20:697-704.
- 68. Brickman AM, Paul RH, Cohen RA, et al. Category and letter verbal fluency across the adult lifespan: relationship to EEG theta power. Arch Clin Neuropsychol 2005;20:561-73.
- 69. Gunstad J, Paul RH, Cohen RA, Tate DF, Spitznagel MB, Gordon E. Elevated body mass index is associated with executive dysfunction in otherwise healthy adults. Compr Psychiatry 2007;48:57-61.
- 70. Koren-Morag N, Goldbourt U, Tanne D. Relation between the metabolic syndrome and ischemic stroke or transient ischemic attack: a prospective cohort study in patients with atherosclerotic cardiovascular disease. Stroke 2005;36:1366-71.
- 71. de la Torre JC. Impaired cerebromicrovascular perfusion. Summary of evidence in support of its causality in Alzheimer's disease. Ann N Y Acad Sci 2000;924:136-52.
- 72. Brown NA, Zenilman ME. The impact of frailty in the elderly on the outcome of surgery in the aged. Advances in surgery 2010;44:229-49.
- 73. Arterburn D, Schauer DP, Wise RE, et al. Change in predicted 10-year cardiovascular risk following laparoscopic Roux-en-Y gastric bypass surgery. Obes Surg 2009;19:184-9.
- 74. Ashrafian H, le Roux CW, Darzi A, Athanasiou T. Effects of bariatric surgery on cardiovascular function. Circulation 2008;118:2091-102.
- 75. Williams KV, Bertoldo A, Kinahan P, Cobelli C, Kelley DE. Weight loss-induced plasticity of glucose transport and phosphorylation in the insulin resistance of obesity and type 2 diabetes. Diabetes 2003;52:1619-26.
- 76. Gunstad J, Strain G, Devlin MJ, et al. Improved memory function 12 weeks after bariatric surgery. Surg Obes Relat Dis 2011;7:465-72.
- 77. Gastrointestinal surgery for severe obesity: National Institutes of Health Consensus Development Conference Statement. The American journal of clinical nutrition 1992;55:615S-9S.
- 78. Santry HP, Gillen DL, Lauderdale DS. Trends in bariatric surgical procedures. JAMA 2005;294:1909-17.
- 79. Buchwald H, Avidor Y, Braunwald E, et al. Bariatric surgery: a systematic review and meta-analysis. JAMA 2004;292:1724-37.
- 80. Colquitt J, Clegg A, Loveman E, Royle P, Sidhu MK. Surgery for morbid obesity. Cochrane database of systematic reviews (Online) 2005:CD003641.
- 81. Maggard MA, Shugarman LR, Suttorp M, et al. Meta-analysis: surgical treatment of obesity. Annals of internal medicine 2005;142:547-59.
- 82. Sjostrom L, Lindroos AK, Peltonen M, et al. Lifestyle, diabetes, and cardiovascular risk factors 10 years after bariatric surgery. The New England journal of medicine 2004;351:2683-93.
- 83. Christou NV, Look D, Maclean LD. Weight gain after short- and long-limb gastric bypass in patients followed for longer than 10 years. Annals of surgery 2006;244:734-40.
- 84. Adams TD, Gress RE, Smith SC, et al. Long-term mortality after gastric bypass surgery. The New England journal of medicine 2007;357:753-61.
- 85. Pories WJ, Swanson MS, MacDonald KG, et al. Who would have thought it? An operation proves to be the most effective therapy for adult-onset diabetes mellitus. Annals of surgery 1995;222:339-50; discussion 50-2.
- 86. Sjostrom L, Narbro K, Sjostrom CD, et al. Effects of bariatric surgery on mortality in Swedish obese subjects. The New England journal of medicine 2007;357:741-52.
- 87. Dixon JB, O'Brien PE, Playfair J, et al. Adjustable gastric banding and conventional therapy for type 2 diabetes: a randomized controlled trial. JAMA 2008;299:316-23.

- 88. Powers KA, Rehrig ST, Jones DB. Financial impact of obesity and bariatric surgery. The Medical clinics of North America 2007;91:321-38, ix.
- 89. Ross MH, Yurgelun-Todd DA, Renshaw PF, et al. Age-related reduction in functional MRI response to photic stimulation. Neurology 1997;48:173-6.
- 90. Schriger DL, Baraff L. Defining normal capillary refill: variation with age, sex, and temperature. Ann Emerg Med 1988;17:932-5.
- 91. Huettel SA, Obembe OO, Song AW, Woldorff MG. The BOLD fMRI refractory effect is specific to stimulus attributes: evidence from a visual motion paradigm. Neuroimage 2004;23:402-8.
- 92. Huettel SA, Singerman JD, McCarthy G. The effects of aging upon the hemodynamic response measured by functional MRI. Neuroimage 2001;13:161-75.
- 93. Taoka T, Iwasaki S, Uchida H, et al. Age correlation of the time lag in signal change on EPI-fMRI. J Comput Assist Tomogr 1998;22:514-7.
- 94. Frodl T, Scheuerecker J, Schoepf V, et al. Different effects of mirtazapine and venlafaxine on brain activation: an open randomized controlled fMRI study. The Journal of clinical psychiatry.
- 95. Lee YS, Han DH, Lee JH, Choi TY. The Effects of Methylphenidate on Neural Substrates Associated with Interference Suppression in Children with ADHD: A Preliminary Study Using Event Related fMRI. Psychiatry investigation;7:49-54.
- 96. Pavuluri MN, Passarotti AM, Parnes SA, Fitzgerald JM, Sweeney JA. A pharmacological functional magnetic resonance imaging study probing the interface of cognitive and emotional brain systems in pediatric bipolar disorder. Journal of child and adolescent psychopharmacology;20:395-406.
- 97. Richter A, Grimm S, Northoff G. Lorazepam modulates orbitofrontal signal changes during emotional processing in catatonia. Human psychopharmacology;25:55-62.
- 98. Bentley P, Driver J, Dolan RJ. Cholinesterase inhibition modulates visual and attentional brain responses in Alzheimer's disease and health. Brain 2008;131:409-24.
- 99. Bryant CA, Jackson SH. Functional imaging of the brain in the evaluation of drug response and its application to the study of aging. Drugs & aging 1998;13:211-22.
- 100. Wierenga CE, Bondi MW. Use of functional magnetic resonance imaging in the early identification of Alzheimer's disease. Neuropsychology review 2007;17:127-43.
- 101. Chaumeil MM, Valette J, Guillermier M, et al. Multimodal neuroimaging provides a highly consistent picture of energy metabolism, validating 31P MRS for measuring brain ATP synthesis. Proceedings of the National Academy of Sciences of the United States of America 2009;106:3988-93.
- 102. Chavez JC, Zaleska MM, Wang X, et al. Multimodal magnetic resonance imaging for assessing evolution of ischemic penumbra: a key translational medicine strategy to manage the risk of developing novel therapies for acute ischemic stroke. J Cereb Blood Flow Metab 2009;29:217-9.
- 103. Haltia LT, Viljanen A, Parkkola R, et al. Brain white matter expansion in human obesity and the recovering effect of dieting. J Clin Endocrinol Metab 2007;92:3278-84.
- 104. Johnson JB, Summer W, Cutler RG, et al. Alternate day calorie restriction improves clinical findings and reduces markers of oxidative stress and inflammation in overweight adults with moderate asthma. Free radical biology & medicine 2007;42:665-74.
- 105. McCaffery JM, Haley AP, Sweet LH, et al. Differential functional magnetic resonance imaging response to food pictures in successful weight-loss maintainers relative to normal-weight and obese controls. The American journal of clinical nutrition 2009;90:928-34.
- 106. DelParigi A, Chen K, Salbe AD, et al. Persistence of abnormal neural responses to a meal in postobese individuals. Int J Obes Relat Metab Disord 2004;28:370-7.
- 107. Le DS, Pannacciulli N, Chen K, et al. Less activation in the left dorsolateral prefrontal cortex in the reanalysis of the response to a meal in obese than in lean women and its association with successful weight loss. The American journal of clinical nutrition 2007;86:573-9.
- 108. Velasco MV, Casanova I, Sanchez-Pernaute A, et al. Unusual late-onset Wernicke's encephalopathy following vertical banded gastroplasty. Obes Surg 2009;19:937-40.

- 109. Aasheim ET. Wernicke encephalopathy after bariatric surgery: a systematic review. Annals of surgery 2008;248:714-20.
- 110. Foster D, Falah M, Kadom N, Mandler R. Wernicke encephalopathy after bariatric surgery: losing more than just weight. Neurology 2005;65:1987; discussion 847.
- 111. Choi JY, Scarborough TK. Stroke and seizure following a recent laparoscopic Roux-en-Y gastric bypass. Obes Surg 2004;14:857-60.
- 112. Loh Y, Watson WD, Verma A, Chang ST, Stocker DJ, Labutta RJ. Acute Wernicke's encephalopathy following bariatric surgery: clinical course and MRI correlation. Obes Surg 2004;14:129-32.
- 113. Mensah GA, Mokdad AH, Ford E, et al. Obesity, metabolic syndrome, and type 2 diabetes: emerging epidemics and their cardiovascular implications. Cardiology clinics 2004;22:485-504.
- 114. Whitmer RA, Gustafson DR, Barrett-Connor E, Haan MN, Gunderson EP, Yaffe K. Central obesity and increased risk of dementia more than three decades later. Neurology 2008;71:1057-64.
- 115. Spies C, Farzaneh-Far R, Na B, Kanaya A, Schiller NB, Whooley MA. Relation of obesity to heart failure hospitalization and cardiovascular events in persons with stable coronary heart disease (from the Heart and Soul Study). Am J Cardiol 2009;104:883-9.
- 116. De Marco M, de Simone G, Roman MJ, et al. Cardiovascular and metabolic predictors of progression of prehypertension into hypertension: the Strong Heart Study. Hypertension 2009;54:974-80.
- 117. Pasquali SK, Marino BS, Pudusseri A, et al. Risk factors and comorbidities associated with obesity in children and adolescents after the arterial switch operation and Ross procedure. American heart journal 2009;158:473-9.
- 118. Dixon JB. The effect of obesity on health outcomes. Molecular and cellular endocrinology 2009.
- 119. Zhou M, Offer A, Yang G, et al. Body mass index, blood pressure, and mortality from stroke: a nationally representative prospective study of 212,000 Chinese men. Stroke 2008;39:753-9.
- 120. Gallego J, Martinez Vila E, Munoz R. Patients at high risk for ischemic stroke: identification and actions. Cerebrovasc Dis 2007;24 Suppl 1:49-63.
- 121. Sacks FM. Metabolic syndrome: epidemiology and consequences. The Journal of clinical psychiatry 2004;65 Suppl 18:3-12.
- 122. Gunstad J, Paul RH, Cohen RA, Tate DF, Gordon E. Obesity is associated with memory deficits in young and middle-aged adults. Eat Weight Disord 2006;11:e15-9.
- 123. McCawley GM, Ferriss JS, Geffel D, Northup CJ, Modesitt SC. Cancer in obese women: potential protective impact of bariatric surgery. Journal of the American College of Surgeons 2009;208:1093-8.
- 124. Merkow RP, Bilimoria KY, McCarter MD, Bentrem DJ. Effect of body mass index on short-term outcomes after collectomy for cancer. Journal of the American College of Surgeons 2009;208:53-61.
- 125. Wang J, Ruotsalainen S, Moilanen L, Lepisto P, Laakso M, Kuusisto J. The metabolic syndrome predicts incident stroke: a 14-year follow-up study in elderly people in Finland. Stroke 2008;39:1078-83.
- 126. Park JH, Kwon HM. Association between metabolic syndrome and previous ischemic lesions in patients with intracranial atherosclerotic stroke. Clinical neurology and neurosurgery 2008;110:215-21.
- 127. Cusi K. Role of obesity and lipotoxicity in the development of nonalcoholic steatohepatitis: pathophysiology and clinical implications. Gastroenterology 2012;142:711-25 e6.
- 128. Lomonaco R, Ortiz-Lopez C, Orsak B, et al. Effect of adipose tissue insulin resistance on metabolic parameters and liver histology in obese patients with nonalcoholic fatty liver disease. Hepatology 2012;55:1389-97.
- 129. Wang S, Kamat A, Pergola P, Swamy A, Tio F, Cusi K. Metabolic factors in the development of hepatic steatosis and altered mitochondrial gene expression *in vivo*. Metabolism 2011;60:1090-9.
- 130. Cusi K. The role of adipose tissue and lipotoxicity in the pathogenesis of type 2 diabetes. Curr Diab Rep 2010;10:306-15.
- 131. Cusi K. Role of insulin resistance and lipotoxicity in non-alcoholic steatohepatitis. Clin Liver Dis 2009;13:545-63.
- 132. Cusi K. Nonalcoholic fatty liver disease in type 2 diabetes mellitus. Curr Opin Endocrinol Diabetes Obes 2009;16:141-9.

- 133. Gastaldelli A, Cusi K, Pettiti M, et al. Relationship between hepatic/visceral fat and hepatic insulin resistance in nondiabetic and type 2 diabetic subjects. Gastroenterology 2007;133:496-506.
- 134. Murdolo G, Smith U. The dysregulated adipose tissue: a connecting link between insulin resistance, type 2 diabetes mellitus and atherosclerosis. Nutr Metab Cardiovasc Dis 2006;16 Suppl 1:S35-8.
- 135. Bugianesi E, Gastaldelli A, Vanni E, et al. Insulin resistance in non-diabetic patients with non-alcoholic fatty liver disease: sites and mechanisms. Diabetologia 2005;48:634-42.
- 136. Harrison SA. Liver disease in patients with diabetes mellitus. J Clin Gastroenterol 2006;40:68-76.
- 137. Choi SS, Diehl AM. Hepatic triglyceride synthesis and nonalcoholic fatty liver disease. Curr Opin Lipidol 2008;19:295-300.
- 138. Choi S, Diehl AM. Role of inflammation in nonalcoholic steatohepatitis. Curr Opin Gastroenterol 2005;21:702-7.
- 139. Gentile CL, Wang D, Pfaffenbach KT, Cox R, Wei Y, Pagliassotti MJ. Fatty acids regulate CREBh via transcriptional mechanisms that are dependent on proteasome activity and insulin. Mol Cell Biochem 2010;344:99-107.
- 140. Gentile CL, Pagliassotti MJ. The role of fatty acids in the development and progression of nonalcoholic fatty liver disease. J Nutr Biochem 2008;19:567-76.
- 141. Kashyap S, Belfort R, Gastaldelli A, et al. A sustained increase in plasma free fatty acids impairs insulin secretion in nondiabetic subjects genetically predisposed to develop type 2 diabetes. Diabetes 2003;52:2461-74.
- 142. Svedberg J, Bjorntorp P, Smith U, Lonnroth P. Effect of free fatty acids on insulin receptor binding and tyrosine kinase activity in hepatocytes isolated from lean and obese rats. Diabetes 1992;41:294-8.
- 143. Svedberg J, Bjorntorp P, Lonnroth P, Smith U. Prevention of inhibitory effect of free fatty acids on insulin binding and action in isolated rat hepatocytes by etomoxir. Diabetes 1991;40:783-6.
- 144. Svedberg J, Bjorntorp P, Smith U, Lonnroth P. Free-fatty acid inhibition of insulin binding, degradation, and action in isolated rat hepatocytes. Diabetes 1990;39:570-4.
- 145. Wiesenthal SR, Sandhu H, McCall RH, et al. Free fatty acids impair hepatic insulin extraction *in vivo*. Diabetes 1999;48:766-74.
- 146. Adiels M, Westerbacka J, Soro-Paavonen A, et al. Acute suppression of VLDL1 secretion rate by insulin is associated with hepatic fat content and insulin resistance. Diabetologia 2007;50:2356-65.
- 147. Luchsinger JA, Mayeux R. Cardiovascular risk factors and Alzheimer's disease. Curr Atheroscler Rep 2004;6:261-6.
- 148. Cereda E, Sacchi MC, Malavazos AE. Central obesity and increased risk of dementia more than three decades later. Neurology 2009;72:1030-1; author reply 1.
- 149. Hughes TF, Borenstein AR, Schofield E, Wu Y, Larson EB. Association between late-life body mass index and dementia: The Kame Project. Neurology 2009;72:1741-6.
- 150. Tezapsidis N, Smith MA, Ashford JW. Central obesity and increased risk of dementia more than three decades later. Neurology 2009;72:1030-1; author reply 1.
- 151. de la Monte SM, Wands JR. Review of insulin and insulin-like growth factor expression, signaling, and malfunction in the central nervous system: relevance to Alzheimer's disease. J Alzheimers Dis 2005;7:45-61.
- 152. Hoyer S. Memory function and brain glucose metabolism. Pharmacopsychiatry 2003;36 Suppl 1:S62-7.
- 153. Rivera EJ, Goldin A, Fulmer N, Tavares R, Wands JR, de la Monte SM. Insulin and insulin-like growth factor expression and function deteriorate with progression of Alzheimer's disease: link to brain reductions in acetylcholine. J Alzheimers Dis 2005;8:247-68.
- 154. Vanhanen M, Soininen H. Glucose intolerance, cognitive impairment and Alzheimer's disease. Curr Opin Neurol 1998;11:673-7.
- 155. Convit A. Links between cognitive impairment in insulin resistance: an explanatory model. Neurobiol Aging 2005;26 Suppl 1:31-5.
- 156. Yaffe K, Blackwell T, Whitmer RA, Krueger K, Barrett Connor E. Glycosylated hemoglobin level and development of mild cognitive impairment or dementia in older women. J Nutr Health Aging 2006;10:293-5.
- 157. Gotkine M. Vascular risk factors and cognitive decline among elderly male twins. Neurology 2007;68:1871; author reply

- 158. Frisardi V, Solfrizzi V, Seripa D, et al. Metabolic-cognitive syndrome: a cross-talk between metabolic syndrome and Alzheimer's disease. Ageing Res Rev;9:399-417.
- 159. Akbaraly TN, Kivimaki M, Shipley MJ, et al. Metabolic syndrome over 10 years and cognitive functioning in late mid life: The Whitehall II study. Diabetes care 2009.
- 160. Alves TC, Busatto GF. Regional cerebral blood flow reductions, heart failure and Alzheimer's disease. Neurol Res 2006;28:579-87.
- 161. Alves TC, Rays J, Fraguas R, Jr., et al. Localized cerebral blood flow reductions in patients with heart failure: a study using 99mTc-HMPAO SPECT. J Neuroimaging 2005;15:150-6.
- 162. Biessels GJ, Kappelle LJ. Increased risk of Alzheimer's disease in Type II diabetes: insulin resistance of the brain or insulin-induced amyloid pathology? Biochem Soc Trans 2005;33:1041-4.
- 163. Weller RO, Cohen NR, Nicoll JA. Cerebrovascular disease and the pathophysiology of Alzheimer's disease. Implications for therapy. Panminerva Med 2004;46:239-51.
- 164. Kalaria RN. The role of cerebral ischemia in Alzheimer's disease. Neurobiol Aging 2000;21:321-30.
- 165. Fleisher AS, Podraza KM, Bangen KJ, et al. Cerebral perfusion and oxygenation differences in Alzheimer's disease risk. Neurobiol Aging 2009;30:1737-48.
- 166. Grammas P, Ovase R. Inflammatory factors are elevated in brain microvessels in Alzheimer's disease. Neurobiol Aging 2001;22:837-42.
- 167. Chong ZZ, Li F, Maiese K. Stress in the brain: novel cellular mechanisms of injury linked to Alzheimer's disease. Brain Res Brain Res Rev 2005;49:1-21.
- 168. Fiala M, Zhang L, Gan X, et al. Amyloid-beta induces chemokine secretion and monocyte migration across a human blood--brain barrier model. Mol Med 1998;4:480-9.
- 169. Hampel H, Haslinger A, Scheloske M, et al. Pattern of interleukin-6 receptor complex immunoreactivity between cortical regions of rapid autopsy normal and Alzheimer's disease brain. Eur Arch Psychiatry Clin Neurosci 2005;255:269-78.
- 170. Tarkowski E. Cytokines in dementias. Curr Drug Targets Inflamm Allergy 2002;1:193-200.
- 171. Droge W, Schipper HM. Oxidative stress and aberrant signaling in aging and cognitive decline. Aging Cell 2007;6:361-70.
- 172. Markesbery WR, Lovell MA. Damage to lipids, proteins, DNA, and RNA in mild cognitive impairment. Arch Neurol 2007;64:954-6.
- 173. Wu A, Ying Z, Gomez-Pinilla F. The interplay between oxidative stress and brain-derived neurotrophic factor modulates the outcome of a saturated fat diet on synaptic plasticity and cognition. Eur J Neurosci 2004;19:1699-707.
- 174. de la Monte SM, Wands JR. Alzheimer's disease is type 3 diabetes-evidence reviewed. Journal of diabetes science and technology 2008;2:1101-13.
- 175. de la Monte SM. Insulin resistance and Alzheimer's disease. BMB reports 2009;42:475-81.
- 176. Fuller JH, Stevens LK, Wang SL. Risk factors for cardiovascular mortality and morbidity: the WHO Mutinational Study of Vascular Disease in Diabetes. Diabetologia 2001;44 Suppl 2:S54-64.
- 177. Mozaffarian D. Trans fatty acids effects on systemic inflammation and endothelial function. Atheroscler Suppl 2006;7:29-32.
- 178. Smith NL, Savage PJ, Heckbert SR, et al. Glucose, blood pressure, and lipid control in older people with and without diabetes mellitus: the Cardiovascular Health Study. J Am Geriatr Soc 2002;50:416-23.
- 179. Tziomalos K, Athyros VG, Karagiannis A, Mikhailidis DP. Endothelial function, arterial stiffness and lipid lowering drugs. Expert Opin Ther Targets 2007;11:1143-60.
- 180. Tilvis RS, Kahonen-Vare MH, Jolkkonen J, Valvanne J, Pitkala KH, Strandberg TE. Predictors of cognitive decline and mortality of aged people over a 10-year period. The journals of gerontology 2004;59:268-74
- 181. Pavlik VN, Hyman DJ, Doody R. Cardiovascular risk factors and cognitive function in adults 30-59 years of age (NHANES III). Neuroepidemiology 2005;24:42-50.
- 182. Nagata K, Sasaki E, Goda K, et al. Cerebrovascular disease in type 2 diabetic patients without hypertension. Stroke 2003;34:e232-3; author reply e-3.

- 183. Ferrucci L, Guralnik JM, Salive ME, et al. Cognitive impairment and risk of stroke in the older population. J Am Geriatr Soc 1996;44:237-41.
- 184. Feil D, Marmon T, Unutzer J. Cognitive impairment, chronic medical illness, and risk of mortality in an elderly cohort. Am J Geriatr Psychiatry 2003;11:551-60.
- 185. Klawans HL, Shekelle RB, Ostfeld AM, Tufo HM. Epidemiology of stroke in elderly persons. Neurology 1970;20:373-4.
- 186. Verhaegen P, Borchelt M, Smith J. Relation between cardiovascular and metabolic disease and cognition in very old age: cross-sectional and longitudinal findings from the berlin aging study. Health Psychol 2003;22:559-69.
- 187. Kernan WN, Inzucchi SE. Type 2 Diabetes Mellitus and Insulin Resistance: Stroke Prevention and Management. Curr Treat Options Neurol 2004;6:443-50.
- 188. Vallbracht KB, Schwimmbeck PL, Seeberg B, Kuhl U, Schultheiss HP. Endothelial dysfunction of peripheral arteries in patients with immunohistologically confirmed myocardial inflammation correlates with endothelial expression of human leukocyte antigens and adhesion molecules in myocardial biopsies. J Am Coll Cardiol 2002;40:515-20.
- 189. Dumont AS, Hyndman ME, Dumont RJ, et al. Improvement of endothelial function in insulin-resistant carotid arteries treated with pravastatin. J Neurosurg 2001;95:466-71.
- 190. Parving HH, Nielsen FS, Bang LE, et al. Macro-microangiopathy and endothelial dysfunction in NIDDM patients with and without diabetic nephropathy. Diabetologia 1996;39:1590-7.
- 191. Woods SC, Seeley RJ, Baskin DG, Schwartz MW. Insulin and the blood-brain barrier. Curr Pharm Des 2003;9:795-800.
- 192. Watson GS, Craft S. Insulin resistance, inflammation, and cognition in Alzheimer's Disease: lessons for multiple sclerosis. J Neurol Sci 2006;245:21-33.
- 193. de la Monte SM, Longato L, Tong M, Wands JR. Insulin resistance and neurodegeneration: roles of obesity, type 2 diabetes mellitus and non-alcoholic steatohepatitis. Curr Opin Investig Drugs 2009;10:1049-60.
- 194. de la Monte SM, Tong M, Lester-Coll N, Plater M, Jr., Wands JR. Therapeutic rescue of neurodegeneration in experimental type 3 diabetes: relevance to Alzheimer's disease. J Alzheimers Dis 2006:10:89-109.
- 195. de la Monte SM, Wands JR. Alzheimer-associated neuronal thread protein mediated cell death is linked to impaired insulin signaling. J Alzheimers Dis 2004;6:231-42.
- 196. de la Monte SM, Wands JR. Molecular indices of oxidative stress and mitochondrial dysfunction occur early and often progress with severity of Alzheimer's disease. J Alzheimers Dis 2006;9:167-81.
- 197. J SR-F, Sa-Roriz TM, Rosset I, et al. (Pre)diabetes, brain aging, and cognition. Biochim Biophys Acta 2009;1792:432-43.
- 198. Swardfager W, Herrmann N, Marzolini S, et al. Brain derived neurotrophic factor, cardiopulmonary fitness and cognition in patients with coronary artery disease. Brain Behav Immun 2011;25:1264-71.
- 199. Thompson D, Pepys MB, Wood SP. The physiological structure of human C-reactive protein and its complex with phosphocholine. Structure 1999;7:169-77.
- 200. Sattar N, Gaw A, Scherbakova O, et al. Metabolic syndrome with and without C-reactive protein as a predictor of coronary heart disease and diabetes in the West of Scotland Coronary Prevention Study. Circulation 2003;108:414-9.
- 201. Wu A, Ying Z, Gomez-Pinilla F. Oxidative stress modulates Sir2alpha in rat hippocampus and cerebral cortex. Eur J Neurosci 2006;23:2573-80.
- 202. Troen AM, Shukitt-Hale B, Chao WH, et al. The cognitive impact of nutritional homocysteinemia in apolipoprotein-E deficient mice. J Alzheimers Dis 2006;9:381-92.
- 203. McNamara RK, Carlson SE. Role of omega-3 fatty acids in brain development and function: potential implications for the pathogenesis and prevention of psychopathology. Prostaglandins Leukot Essent Fatty Acids 2006;75:329-49.
- 204. Matsui T, Nemoto M, Maruyama M, et al. Plasma homocysteine and risk of coexisting silent brain infarction in Alzheimer's disease. Neurodegener Dis 2005;2:299-304.

- 205. Markesbery WR, Kryscio RJ, Lovell MA, Morrow JD. Lipid peroxidation is an early event in the brain in amnestic mild cognitive impairment. Ann Neurol 2005;58:730-5.
- 206. Dik MG, Jonker C, Hack CE, Smit JH, Comijs HC, Eikelenboom P. Serum inflammatory proteins and cognitive decline in older persons. Neurology 2005;64:1371-7.
- 207. Galimberti D, Fenoglio C, Lovati C, et al. Serum MCP-1 levels are increased in mild cognitive impairment and mild Alzheimer's disease. Neurobiol Aging 2006;27:1763-8.
- 208. Galimberti D, Schoonenboom N, Scheltens P, et al. Intrathecal chemokine levels in Alzheimer disease and frontotemporal lobar degeneration. Neurology 2006;66:146-7.
- 209. Lindberg C, Chromek M, Ahrengart L, Brauner A, Schultzberg M, Garlind A. Soluble interleukin-1 receptor type II, IL-18 and caspase-1 in mild cognitive impairment and severe Alzheimer's disease. Neurochemistry international 2005;46:551-7.
- 210. Todd Roach J, Volmar CH, Dwivedi S, et al. Behavioral effects of CD40-CD40L pathway disruption in aged PSAPP mice. Brain research 2004;1015:161-8.
- 211. Sun L, Gao YH, Tian DK, et al. Inflammation of different tissues in spontaneously hypertensive rats. Sheng Li Xue Bao 2006;58:318-23.
- 212. Guzik TJ, Mangalat D, Korbut R. Adipocytokines novel link between inflammation and vascular function? J Physiol Pharmacol 2006;57:505-28.
- 213. Bruunsgaard H. Effects of tumor necrosis factor-alpha and interleukin-6 in elderly populations. Eur Cytokine Netw 2002;13:389-91.
- 214. Das UN. Beneficial effect(s) of n-3 fatty acids in cardiovascular diseases: but, why and how? Prostaglandins Leukot Essent Fatty Acids 2000;63:351-62.
- 215. Krabbe KS, Pedersen M, Bruunsgaard H. Inflammatory mediators in the elderly. Experimental gerontology 2004;39:687-99.
- 216. Sun YX, Minthon L, Wallmark A, Warkentin S, Blennow K, Janciauskiene S. Inflammatory markers in matched plasma and cerebrospinal fluid from patients with Alzheimer's disease. Dement Geriatr Cogn Disord 2003;16:136-44.
- 217. Hoth KF, Haley AP, Gunstad J, et al. Elevated C-reactive protein is related to cognitive decline in older adults with cardiovascular disease. J Am Geriatr Soc 2008;56:1898-903.
- 218. Gunstad J, Benitez A, Hoth KF, et al. P-Selectin 1087G/A Polymorphism Is Associated With Neuropsychological Test Performance in Older Adults With Cardiovascular Disease. Stroke 2009.
- 219. Gunstad J, Bausserman L, Paul RH, et al. C-reactive protein, but not homocysteine, is related to cognitive dysfunction in older adults with cardiovascular disease. J Clin Neurosci 2006;13:540-6.
- 220. Cohen R, Gongvantana A, Tashima K, Navia B. . Attention and executive function impairments associated with cytokine Journal of Neuroimmunology In press.
- 221. Rafnsson SB, Deary IJ, Smith FB, et al. Cognitive decline and markers of inflammation and hemostasis: the Edinburgh Artery Study. J Am Geriatr Soc 2007;55:700-7.
- 222. Marioni RE, Strachan MW, Reynolds RM, et al. Association between raised inflammatory markers and cognitive decline in elderly people with type 2 diabetes: the Edinburgh Type 2 Diabetes Study. Diabetes 2010;59:710-3.
- 223. Vallejo AN, Hamel DL, Jr., Mueller RG, et al. NK-like T cells and plasma cytokines, but not anti-viral serology, define immune fingerprints of resilience and mild disability in exceptional aging. PLoS One 2011;6:e26558.
- 224. Villeda SA, Luo J, Mosher KI, et al. The ageing systemic milieu negatively regulates neurogenesis and cognitive function. Nature 2011;477:90-4.
- 225. Gunstad J, Spitznagel MB, Keary TA, et al. Serum leptin levels are associated with cognitive function in older adults. Brain research 2008;1230:233-6.
- 226. Holden KF, Lindquist K, Tylavsky FA, Rosano C, Harris TB, Yaffe K. Serum leptin level and cognition in the elderly: Findings from the Health ABC Study. Neurobiol Aging 2009;30:1483-9.
- 227. Warren MW, Hynan LS, Weiner MF. Leptin and cognition. Dement Geriatr Cogn Disord 2012;33:410-5.

- 228. Warren MW, Hynan LS, Weiner MF. Lipids and adipokines as risk factors for Alzheimer's disease. J Alzheimers Dis 2012;29:151-7.
- 229. Corsi MM, Licastro F, Porcellini E, et al. Reduced plasma levels of P-selectin and L-selectin in a pilot study from Alzheimer disease: relationship with neuro-degeneration. Biogerontology 2011;12:451-4.
- 230. Martinez-Cengotitabengoa M, Mac-Dowell KS, Leza JC, et al. Cognitive impairment is related to oxidative stress and chemokine levels in first psychotic episodes. Schizophr Res 2012;137:66-72.
- 231. Moser DJ, Cohen RA, Clark MM, et al. Neuropsychological functioning among cardiac rehabilitation patients. J Cardiopulm Rehabil 1999;19:91-7.
- 232. Browndyke JN, Moser DJ, Cohen RA, et al. Acute neuropsychological functioning following cardiosurgical interventions associated with the production of intraoperative cerebral microemboli. Clin Neuropsychol 2002;16:463-71.
- 233. Gunstad J, Macgregor KL, Paul RH, et al. Cardiac rehabilitation improves cognitive performance in older adults with cardiovascular disease. J Cardiopulm Rehabil 2005;25:173-6.
- 234. Gunstad J, Cohen RA, Paul RH, Tate DF, Hoth KF, Poppas A. Understanding reported cognitive dysfunction in older adults with cardiovascular disease. Neuropsychiatr Dis Treat 2006;2:213-8.
- 235. Gunstad J, Paul RH, Brickman AM, et al. Patterns of cognitive performance in middle-aged and older adults: A cluster analytic examination. J Geriatr Psychiatry Neurol 2006;19:59-64.
- 236. Gunstad J, Poppas A, Smeal S, et al. Relation of brain natriuretic peptide levels to cognitive dysfunction in adults > 55 years of age with cardiovascular disease. Am J Cardiol 2006;98:538-40.
- 237. Haley AP, Sweet LH, Gunstad J, et al. Verbal working memory and atherosclerosis in patients with cardiovascular disease: an fMRI study. J Neuroimaging 2007;17:227-33.
- 238. Keary TA, Gunstad J, Poppas A, et al. Blood pressure variability and dementia rating scale performance in older adults with cardiovascular disease. Cogn Behav Neurol 2007;20:73-7.
- 239. Forman DE, Cohen R.A., Hoth K.F., Haley A.P., Poppas A., Moser D.J., Gunstad J., Gerhard-Herman M. Vascular health and cognitive function in older adults with cardiovascular disease. Artery Research 2008;2 (1), pp.: 35-43.
- 240. Hoth K, Poppas A, Moser DJ, Paul RH, Cohen RA. . Cardiac dysfunction and cognition in older adults with heart failure. Cogn Behav Neurol 2008;21:65-72.
- 241. Haley AP, Hoth KF, Gunstad J, et al. Subjective cognitive complaints relate to white matter hyperintensities and future cognitive decline in patients with cardiovascular disease. Am J Geriatr Psychiatry 2009;17:976-85.
- 242. Irani F, Sweet LH, Haley AP, Gunstad JJ, Jerskey BA, Mulligan RC, Jefferson AL, Poppas A, Cohen RA1. A fMRI Study of Verbal Working Memory, Cardiac Output, and Ejection Fraction in Elderly Patients with Cardiovascular Disease Brain Imaging Behav 2009;3:350-7.
- 243. Jerskey BA, Cohen RA, Jefferson AL, et al. Sustained attention is associated with left ventricular ejection fraction in older adults with heart disease. J Int Neuropsychol Soc 2009;15:137-41.
- 244. Hoth KF, Poppas A, Ellison KE, et al. Link Between Change in Cognition and Left Ventricular Function Following Cardiac Resynchronization Therapy. Journal of cardiopulmonary rehabilitation and prevention 2010.
- 245. Okonkwo OC, Cohen RA Gunstad J, Tremont G, Alosco ML, Poppas A. Longitudinal trajectories of cognitive decline among older adults with cardiovascular disease Cerebrovascular Disease 2010.
- 246. Berzin TM, Zipser BD, Rafii MS, et al. Agrin and microvascular damage in Alzheimer's disease. Neurobiol Aging 2000;21:349-55.
- 247. Farkas E, De Vos RA, Jansen Steur EN, Luiten PG. Are Alzheimer's disease, hypertension, and cerebrocapillary damage related? Neurobiol Aging 2000;21:235-43.
- 248. Miao J, Vitek MP, Xu F, Previti ML, Davis J, Van Nostrand WE. Reducing cerebral microvascular amyloid-beta protein deposition diminishes regional neuroinflammation in vasculotropic mutant amyloid precursor protein transgenic mice. J Neurosci 2005;25:6271-7.
- 249. Claudio L. Ultrastructural features of the blood-brain barrier in biopsy tissue from Alzheimer's disease patients. Acta Neuropathol (Berl) 1996;91:6-14.

- 250. Folin M, Baiguera S, Tommasini M, et al. Effects of beta-amyloid on rat neuromicrovascular endothelial cells cultured in vitro. Int J Mol Med 2005;15:929-35.
- 251. Khalil Z, Chen H, Helme RD. Mechanisms underlying the vascular activity of beta-amyloid protein fragment (beta A(4)25-35) at the level of skin microvasculature. Brain research 1996;736:206-16.
- 252. Ravi LB, Mohanty JG, Chrest FJ, et al. Influence of beta-amyloid fibrils on the interactions between red blood cells and endothelial cells. Neurol Res 2004;26:579-85.
- 253. Salloway S, Gur T, Berzin T, et al. Effect of APOE genotype on microvascular basement membrane in Alzheimer's disease. J Neurol Sci 2002;203-204:183-7.
- 254. Zipser BD, Johanson CE, Gonzalez L, et al. Microvascular injury and blood-brain barrier leakage in Alzheimer's disease. Neurobiol Aging 2006.
- 255. Acanfora D, Trojano L, Iannuzzi GI, et al. The brain in congestive heart failure. Arch Gerontol Geriatr 1996;23:247-56.
- 256. Almeida OP, Flicker L. The mind of a failing heart: a systematic review of the association between congestive heart failure and cognitive functioning. Internal Medicine Journal 2001;31:290-5.
- 257. Alves TC, Rays J, Fraguas R, Jr., et al. Localized cerebral blood flow reductions in patients with heart failure: a study using 99mTc-HMPAO SPECT. Journal of Neuroimaging 2005;15:150-6.
- 258. Bowler JV, Steenhuis R, Hachinski V. Conceptual background to vascular cognitive impairment. Alzheimer Dis Assoc Disord 1999;13 Suppl 3:S30-7.
- 259. Claus JJ, Breteler MM, Hasan D, et al. Vascular risk factors, atherosclerosis, cerebral white matter lesions and cerebral perfusion in a population-based study. Eur J Nucl Med 1996;23:675-82.
- 260. Cohen RA, Poppas A, Forman D, et al. Vascular and Cognitive Functions Associated with Cardiovascular Disease in the Elderly. Journal of Clinical and Experimental Neuropsychology 2009:1-15.
- 261. de Leeuw FE, Richard F, de Groot JC, et al. Interaction between hypertension, apoE, and cerebral white matter lesions. Stroke 2004;35:1057-60.
- 262. Firbank MJ, Wiseman RM, Burton EJ, Saxby BK, O'Brien JT, Ford GA. Brain atrophy and white matter hyperintensity change in older adults and relationship to blood pressure. Brain atrophy, WMH change and blood pressure. Journal of neurology 2007;254:713-21.
- 263. Geroldi C, Ferrucci L, Bandinelli S, et al. Mild cognitive deterioration with subcortical features: prevalence, clinical characteristics, and association with cardiovascular risk factors in community-dwelling older persons (The InCHIANTI Study). J Am Geriatr Soc 2003;51:1064-71.
- 264. Jefferson AL, Poppas A, Paul RH, Cohen RA. Systemic hypoperfusion is associated with executive dysfunction in geriatric cardiac patients. Neurobiol Aging 2007;28:477-83.
- 265. Moser DJ, Hoth KF, Robinson RG, et al. Blood vessel function and cognition in elderly patients with atherosclerosis. Stroke 2004;35:e369-72.
- 266. Vogels RL, Oosterman JM, van Harten B, et al. Profile of cognitive impairment in chronic heart failure. Journal of the American Geriatrics Society 2007;55:1764-70.
- 267. Guo Z, Viitanen M, Winblad B, Fratiglioni L. Low blood pressure and incidence of dementia in a very old sample: dependent on initial cognition. J Am Geriatr Soc 1999;47:723-6.
- 268. Okonkwo OC, Cohen RA, Gunstad J, Poppas A. Cardiac output, blood pressure variability, and cognitive decline in geriatric cardiac patients. Journal of cardiopulmonary rehabilitation and prevention 2011;31:290-7.
- 269. Kristensen PL, Hoi-Hansen T, Boomsma F, Pedersen-Bjergaard U, Thorsteinsson B. Vascular endothelial growth factor during hypoglycemia in patients with type 1 diabetes mellitus: relation to cognitive function and renin-angiotensin system activity. Metabolism 2009;58:1430-8.
- 270. Huber JD. Diabetes, cognitive function, and the blood-brain barrier. Curr Pharm Des 2008;14:1594-600.
- 271. Wang Y, Galvan V, Gorostiza O, Ataie M, Jin K, Greenberg DA. Vascular endothelial growth factor improves recovery of sensorimotor and cognitive deficits after focal cerebral ischemia in the rat. Brain research 2006;1115:186-93.
- 272. de la Torre JC, Aliev G. Inhibition of vascular nitric oxide after rat chronic brain hypoperfusion: spatial memory and immunocytochemical changes. J Cereb Blood Flow Metab 2005;25:663-72.

- 273. Stanek KM, Gunstad J, Paul RH, et al. Longitudinal cognitive performance in older adults with cardiovascular disease: evidence for improvement in heart failure. J Cardiovasc Nurs 2009;24:192-7.
- 274. Knopman DS. Cerebrovascular disease and dementia. The British journal of radiology 2007;80 Spec No 2:S121-7.
- 275. Pereira AA, Weiner DE, Scott T, et al. Subcortical cognitive impairment in dialysis patients. Hemodialysis international 2007;11:309-14.
- 276. Vidal JS, Sigurdsson S, Jonsdottir MK, et al. Coronary artery calcium, brain function and structure: the AGES-Reykjavik Study. Stroke 2010;41:891-7.
- 277. Vinkers DJ, Stek ML, van der Mast RC, et al. Generalized atherosclerosis, cognitive decline, and depressive symptoms in old age. Neurology 2005;65:107-12.
- 278. Beebe DW, Groesz L, Wells C, Nichols A, McGee K. The neuropsychological effects of obstructive sleep apnea: a meta-analysis of norm-referenced and case-controlled data. Sleep 2003;26:298-307.
- 279. Bédard M-A, Montplaisir J, Richer F, Rouleau I, Malo J. Obstructive Sleep Apnea Syndrome: Pathogenesis of Neuropsychological Deficits. Journal of Clinical and Experimental Neuropsychology 1991;13:950-64.
- 280. Naegele B, Thouvard V, Pepin JL, et al. Deficits of cognitive executive functions in patients with sleep apnea syndrome. Sleep 1995;18:43-52.
- 281. Roehrs T, Merrion M, Pedrosi B, Stepanski E, Zorick F, Roth T. Neuropsychological function in obstructive sleep apnea syndrome (OSAS) compared to chronic obstructive pulmonary disease (COPD). Sleep 1995;18:382-8.
- 282. Beebe DW, Gozal D. Obstructive sleep apnea and the prefrontal cortex: towards a comprehensive model linking nocturnal upper airway obstruction to daytime cognitive and behavioral deficits. Journal of Sleep Research 2002;11:1-16.
- 283. Morgenthaler TI, Aurora RN, Brown T, et al. Practice parameters for the use of autotitrating continuous positive airway pressure devices for titrating pressures and treating adult patients with obstructive sleep apnea syndrome: an update for 2007. An American Academy of Sleep Medicine report. Sleep 2008;31:141-7.
- 284. Kushida CA, Littner MR, Hirshkowitz M, et al. Practice parameters for the use of continuous and bilevel positive airway pressure devices to treat adult patients with sleep-related breathing disorders. Sleep 2006;29:375-80.
- 285. Kylstra WA, Aaronson JA, Hofman WF, Schmand BA. Neuropsychological functioning after CPAP treatment in obstructive sleep apnea: A meta-analysis. Sleep medicine reviews 2012.
- 286. Castriotta RJ, Wilde MC, Lai JM, Atanasov S, Masel BE, Kuna ST. Prevalence and consequences of sleep disorders in traumatic brain injury. J Clin Sleep Med 2007;3:349-56.
- 287. Ohayon MM, Vecchierini MF. Normative sleep data, cognitive function and daily living activities in older adults in the community. Sleep 2005;28:981-9.
- 288. Sateia MJ. Neuropsychological impairment and quality of life in obstructive sleep apnea. Clin Chest Med 2003;24:249-59.
- 289. Boeka AG, Lokken KL. Neuropsychological performance of a clinical sample of extremely obese individuals. Arch Clin Neuropsychol 2008;23:467-74.
- 290. Almeida JR, Versace A, Mechelli A, et al. Abnormal amygdala-prefrontal effective connectivity to happy faces differentiates bipolar from major depression. Biol Psychiatry 2009;66:451-9.
- 291. Boldrini M, Hen R, Underwood MD, et al. Hippocampal angiogenesis and progenitor cell proliferation are increased with antidepressant use in major depression. Biol Psychiatry 2012;72:562-71.
- 292. Chantiluke K, Halari R, Simic M, et al. Fronto-striato-cerebellar dysregulation in adolescents with depression during motivated attention. Biol Psychiatry 2012;71:59-67.
- 293. Cole J, Chaddock CA, Farmer AE, et al. White matter abnormalities and illness severity in major depressive disorder. Br J Psychiatry 2012;201:33-9.
- 294. Juhasz G, Dunham JS, McKie S, et al. The CREB1-BDNF-NTRK2 pathway in depression: multiple gene-cognition-environment interactions. Biol Psychiatry 2011;69:762-71.

- 295. Cohen R, Lohr I, Paul R, Boland R. Impairments of attention and effort among patients with major affective disorders. J Neuropsychiatry Clin Neurosci 2001;13:385-95.
- 296. Byrne ML, Sheeber L, Simmons JG, et al. Autonomic cardiac control in depressed adolescents. Depress Anxiety 2010;27:1050-6.
- 297. Hach I, Ruhl UE, Klose M, Klotsche J, Kirch W, Jacobi F. Obesity and the risk for mental disorders in a representative German adult sample. Eur J Public Health 2007;17:297-305.
- 298. Hach I, Ruhl UE, Klotsche J, Klose M, Jacobi F. Associations between waist circumference and depressive disorders. J Affect Disord 2006;92:305-8.
- 299. Pessina A, Andreoli M, Vassallo C. Adaptability and compliance of the obese patient to restrictive gastric surgery in the short term. Obes Surg 2001;11:459-63.
- 300. Zimmerman M, Hrabosky JI, Francione C, et al. Impact of obesity on the psychometric properties of the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition criteria for major depressive disorder. Compr Psychiatry 2011;52:146-50.
- 301. Sweet LH, Hassenstab JJ, McCaffery JM, et al. Brain response to food stimulation in obese, normal weight, and successful weight loss maintainers. Obesity (Silver Spring) 2012;20:2220-5.
- 302. Di Bello V, Santini F, Di Cori A, et al. Effects of bariatric surgery on early myocardial alterations in adult severely obese subjects. Cardiology 2008;109:241-8.
- 303. Randall OS, Kwagyan J, Huang Z, Xu S, Ketete M, Maqbool AR. Effect of diet and exercise on pulse pressure and cardiac function in morbid obesity: analysis of 24-hour ambulatory blood pressure. Journal of clinical hypertension (Greenwich, Conn 2005;7:455-63.
- 304. Cohen RV, Pinheiro JC, Schiavon CA, Salles JE, Wajchenberg BL, Cummings DE. Effects of gastric bypass surgery in patients with type 2 diabetes and only mild obesity. Diabetes care 2012;35:1420-8.
- 305. Pepperell JC. Sleep apnoea syndromes and the cardiovascular system. Clin Med 2011;11:275-8.
- 306. Shah SS, Todkar JS, Shah PS, Cummings DE. Diabetes remission and reduced cardiovascular risk after gastric bypass in Asian Indians with body mass index <35 kg/m(2). Surg Obes Relat Dis 2010;6:332-8.
- 307. Buchwald H, Estok R, Fahrbach K, et al. Weight and type 2 diabetes after bariatric surgery: systematic review and meta-analysis. The American journal of medicine 2009;122:248-56 e5.
- 308. Hussain A, Mahmood H, El-Hasani S. Can Roux-en-Y gastric bypass provide a lifelong solution for diabetes mellitus? Canadian journal of surgery 2009;52:E269-75.
- 309. Kadera BE, Lum K, Grant J, Pryor AD, Portenier DD, DeMaria EJ. Remission of type 2 diabetes after Roux-en-Y gastric bypass is associated with greater weight loss. Surg Obes Relat Dis 2009;5:305-9.
- 310. Simon I, Escote X, Vilarrasa N, et al. Adipocyte fatty acid-binding protein as a determinant of insulin sensitivity in morbid-obese women. Obesity (Silver Spring) 2009;17:1124-8.
- 311. Trakhtenbroit MA, Leichman JG, Algahim MF, et al. Body weight, insulin resistance, and serum adipokine levels 2 years after 2 types of bariatric surgery. The American journal of medicine 2009;122:435-42.
- 312. Vila M, Ruiz O, Belmonte M, et al. Changes in lipid profile and insulin resistance in obese patients after Scopinaro biliopancreatic diversion. Obes Surg 2009;19:299-306.
- 313. Shah PS, Todkar JS, Shah SS. Effectiveness of laparoscopic sleeve gastrectomy on glycemic control in obese Indians with type 2 diabetes mellitus. Surg Obes Relat Dis 2010;6:138-41.
- 314. Pournaras DJ, Osborne A, Hawkins SC, et al. Remission of type 2 diabetes after gastric bypass and banding: mechanisms and 2 year outcomes. Annals of surgery 2010;252:966-71.
- 315. O'Brien PE. Bariatric surgery: mechanisms, indications and outcomes. J Gastroenterol Hepatol 2010:25:1358-65.
- 316. Caiazzo R, Arnalsteen L, Pigeyre M, et al. Long-term metabolic outcome and quality of life after laparoscopic adjustable gastric banding in obese patients with type 2 diabetes mellitus or impaired fasting glucose. Br J Surg 2010;97:884-91.
- 317. Wang Y, Zhang C. Bariatric Surgery to Correct Morbid Obesity Also Ameliorates Atherosclerosis in Patients with Type 2 Diabetes Mellitus. American journal of biomedical sciences 2009;1:56-69.
- 318. Habib P, Scrocco JD, Terek M, Vanek V, Mikolich JR. Effects of bariatric surgery on inflammatory, functional and structural markers of coronary atherosclerosis. Am J Cardiol 2009;104:1251-5.

- 319. Sturm W, Tschoner A, Engl J, et al. Effect of bariatric surgery on both functional and structural measures of premature atherosclerosis. European heart journal 2009;30:2038-43.
- 320. Sarmento PL, Plavnik FL, Zanella MT, Pinto PE, Miranda RB, Ajzen SA. Association of carotid intimamedia thickness and cardiovascular risk factors in women pre- and post-bariatric surgery. Obes Surg 2009;19:339-44.
- 321. Hofso D, Nordstrand N, Johnson LK, et al. Obesity-related cardiovascular risk factors after weight loss: a clinical trial comparing gastric bypass surgery and intensive lifestyle intervention. Eur J Endocrinol 2010;163:735-45.
- 322. Zambon S, Romanato G, Sartore G, et al. Bariatric surgery improves atherogenic LDL profile by triglyceride reduction. Obes Surg 2009;19:190-5.
- 323. Guajardo-Salinas GE, Hilmy A, Martinez-Ugarte ML. Predictors of weight loss and effectiveness of Rouxen-Y gastric bypass in the morbidly obese Hispano-American population. Obes Surg 2008;18:1369-75.
- 324. Serpa Neto A, Bianco Rossi FM, Dal Moro Amarante R, Alves Buriti N, Cunha Barbosa Saheb G, Rossi M. Effect of weight loss after Roux-en-Y gastric bypass, on renal function and blood pressure in morbidly obese patients. Journal of nephrology 2009;22:637-46.
- 325. de Freitas AC, Campos AC, Coelho JC. The impact of bariatric surgery on nonalcoholic fatty liver disease. Current opinion in clinical nutrition and metabolic care 2008;11:267-74.
- 326. Heath ML, Kow L, Slavotinek JP, Valentine R, Toouli J, Thompson CH. Abdominal adiposity and liver fat content 3 and 12 months after gastric banding surgery. Metabolism 2009;58:753-8.
- 327. Lam BP, Younossi ZM. Treatment regimens for non-alcoholic fatty liver disease. Ann Hepatol 2009;8 Suppl 1:S51-9.
- 328. Mathurin P, Hollebecque A, Arnalsteen L, et al. Prospective study of the long-term effects of bariatric surgery on liver injury in patients without advanced disease. Gastroenterology 2009;137:532-40.
- 329. Mummadi RR, Kasturi KS, Chennareddygari S, Sood GK. Effect of bariatric surgery on nonalcoholic fatty liver disease: systematic review and meta-analysis. Clin Gastroenterol Hepatol 2008;6:1396-402.
- 330. Riedl M, Vila G, Maier C, et al. Plasma osteopontin increases after bariatric surgery and correlates with markers of bone turnover but not with insulin resistance. J Clin Endocrinol Metab 2008;93:2307-12.
- 331. Schaller G, Aso Y, Schernthaner GH, et al. Increase of osteopontin plasma concentrations after bariatric surgery independent from inflammation and insulin resistance. Obes Surg 2009;19:351-6.
- 332. Vasudevan AR, Wu H, Xydakis AM, et al. Eotaxin and obesity. J Clin Endocrinol Metab 2006;91:256-61.
- 333. Bangen KJ, Restom K, Liu TT, et al. Differential age effects on cerebral blood flow and BOLD response to encoding: associations with cognition and stroke risk. Neurobiol Aging 2009;30:1276-87.
- 334. Restom K, Bangen KJ, Bondi MW, Perthen JE, Liu TT. Cerebral blood flow and BOLD responses to a memory encoding task: a comparison between healthy young and elderly adults. Neuroimage 2007;37:430-9.
- 335. Alsop DC, Casement M, de Bazelaire C, Fong T, Press DZ. Hippocampal hyperperfusion in Alzheimer's disease. Neuroimage 2008;42:1267-74.
- 336. Basso M, Yang J, Warren L, et al. Volumetry of amygdala and hippocampus and memory performance in Alzheimer's disease. Psychiatry research 2006;146:251-61.
- 337. Dickerson BC, Salat DH, Greve DN, et al. Increased hippocampal activation in mild cognitive impairment compared to normal aging and AD. Neurology 2005;65:404-11.
- 338. Eidelberg D. Metabolic brain networks in neurodegenerative disorders: a functional imaging approach. Trends in neurosciences 2009;32:548-57.
- 339. Krishnan S, Talley BD, Slavin MJ, Doraiswamy PM, Petrella JR. Current status of functional MR imaging, perfusion-weighted imaging, and diffusion-tensor imaging in Alzheimer's disease diagnosis and research. Neuroimaging clinics of North America 2005;15:853-68, xi.
- 340. Masdeu JC, Zubieta JL, Arbizu J. Neuroimaging as a marker of the onset and progression of Alzheimer's disease. J Neurol Sci 2005;236:55-64.
- 341. Matsuda H. The role of neuroimaging in mild cognitive impairment. Neuropathology 2007;27:570-7.
- 342. Minati L, Grisoli M, Bruzzone MG. MR spectroscopy, functional MRI, and diffusion-tensor imaging in the aging brain: a conceptual review. J Geriatr Psychiatry Neurol 2007;20:3-21.

- 343. Mondadori CR, Buchmann A, Mustovic H, et al. Enhanced brain activity may precede the diagnosis of Alzheimer's disease by 30 years. Brain 2006;129:2908-22.
- 344. Prvulovic D, Van de Ven V, Sack AT, Maurer K, Linden DE. Functional activation imaging in aging and dementia. Psychiatry research 2005;140:97-113.
- 345. Sole-Padulles C, Bartres-Faz D, Junque C, et al. Brain structure and function related to cognitive reserve variables in normal aging, mild cognitive impairment and Alzheimer's disease. Neurobiol Aging 2009;30:1114-24.
- 346. Sperling R. Functional MRI studies of associative encoding in normal aging, mild cognitive impairment, and Alzheimer's disease. Ann N Y Acad Sci 2007;1097:146-55.
- 347. Wang H, Golob EJ, Su MY. Vascular volume and blood-brain barrier permeability measured by dynamic contrast enhanced MRI in hippocampus and cerebellum of patients with MCI and normal controls. J Magn Reson Imaging 2006;24:695-700.
- 348. Yetkin FZ, Rosenberg RN, Weiner MF, Purdy PD, Cullum CM. FMRI of working memory in patients with mild cognitive impairment and probable Alzheimer's disease. European radiology 2006;16:193-206.
- 349. Detre JA, Alsop DC. Perfusion magnetic resonance imaging with continuous arterial spin labeling: methods and clinical applications in the central nervous system. European journal of radiology 1999;30:115-24.
- 350. Dai W, Lopez OL, Carmichael OT, Becker JT, Kuller LH, Gach HM. Abnormal regional cerebral blood flow in cognitively normal elderly subjects with hypertension. Stroke 2008;39:349-54.
- 351. Beason-Held LL, Moghekar A, Zonderman AB, Kraut MA, Resnick SM. Longitudinal changes in cerebral blood flow in the older hypertensive brain. Stroke 2007;38:1766-73.
- 352. Lee CW, Lee JH, Kim JJ, et al. Cerebral metabolic abnormalities in congestive heart failure detected by proton magnetic resonance spectroscopy. J Am Coll Cardiol 1999;33:1196-202.
- 353. Lee CW, Lee JH, Lim TH, et al. Prognostic significance of cerebral metabolic abnormalities in patients with congestive heart failure. Circulation 2001;103:2784-7.
- 354. Lee CW, Lee JH, Yang HS, et al. Effects of heart transplantation on cerebral metabolic abnormalities in patients with congestive heart failure. J Heart Lung Transplant 2006;25:353-5.
- 355. Malloy CR. Correlation of cerebral metabolites with clinical outcome among patients with severe congestive heart failure. Circulation 2001;103:2771-2.
- 356. Lyoo IK, Yoon SJ, Musen G, et al. Altered prefrontal glutamate-glutamine-gamma-aminobutyric acid levels and relation to low cognitive performance and depressive symptoms in type 1 diabetes mellitus. Archives of general psychiatry 2009;66:878-87.
- 357. Haroon E, Watari K, Thomas A, et al. Prefrontal myo-inositol concentration and visuospatial functioning among diabetic depressed patients. Psychiatry research 2009;171:10-9.
- 358. Heikkila O, Lundbom N, Timonen M, Groop PH, Heikkinen S, Makimattila S. Risk for metabolic syndrome predisposes to alterations in the thalamic metabolism. Metabolic brain disease 2008;23:315-24.
- 359. Cherubini A, Luccichenti G, Peran P, et al. Multimodal fMRI tractography in normal subjects and in clinically recovered traumatic brain injury patients. Neuroimage 2007;34:1331-41.
- 360. Gerstl F, Windischberger C, Mitterhauser M, et al. Multimodal imaging of human early visual cortex by combining functional and molecular measurements with fMRI and PET. Neuroimage 2008;41:204-11.
- 361. Walhovd KB, Fjell AM, Amlien I, et al. Multimodal imaging in mild cognitive impairment: Metabolism, morphometry and diffusion of the temporal-parietal memory network. Neuroimage 2009;45:215-23.
- 362. Guye M, Parker GJ, Symms M, et al. Combined functional MRI and tractography to demonstrate the connectivity of the human primary motor cortex *in vivo*. Neuroimage 2003;19:1349-60.
- 363. Haley A, Gunstad JJ, Cohen RA, Jerskey BA, Mulligan RC, Sweet LH. . 2008, . Neural Correlates of Visuospatial Working Memory in Healthy Young Adults at Risk for Hypertension. Brain Imaging and Behavior 2008;2: 192-9.
- 364. Martin LE, Holsen LM, Chambers RJ, et al. Neural mechanisms associated with food motivation in obese and healthy weight adults. Obesity (Silver Spring);18:254-60.

- 365. Passamonti L, Rowe JB, Schwarzbauer C, Ewbank MP, von dem Hagen E, Calder AJ. Personality predicts the brain's response to viewing appetizing foods: the neural basis of a risk factor for overeating. J Neurosci 2009;29:43-51.
- 366. Porubska K, Veit R, Preissl H, Fritsche A, Birbaumer N. Subjective feeling of appetite modulates brain activity: an fMRI study. Neuroimage 2006;32:1273-80.
- 367. Rothemund Y, Preuschhof C, Bohner G, et al. Differential activation of the dorsal striatum by high-calorie visual food stimuli in obese individuals. Neuroimage 2007;37:410-21.
- 368. Stice E, Spoor S, Bohon C, Veldhuizen MG, Small DM. Relation of reward from food intake and anticipated food intake to obesity: a functional magnetic resonance imaging study. Journal of abnormal psychology 2008;117:924-35.
- 369. Stoeckel LE, Kim J, Weller RE, Cox JE, Cook EW, 3rd, Horwitz B. Effective connectivity of a reward network in obese women. Brain research bulletin 2009;79:388-95.
- 370. Brody AL, Mandelkern MA, Jarvik ME, et al. Differences between smokers and nonsmokers in regional gray matter volumes and densities. Biol Psychiatry 2004;55:77-84.
- 371. David SP, Munafo MR, Johansen-Berg H, et al. Effects of Acute Nicotine Abstinence on Cue-elicited Ventral Striatum/Nucleus Accumbens Activation in Female Cigarette Smokers: A Functional Magnetic Resonance Imaging Study. Brain Imaging Behav 2007;1:43-57.
- 372. Bang OY. Multimodal MRI for ischemic stroke: from acute therapy to preventive strategies. Journal of clinical neurology (Seoul, Korea) 2009;5:107-19.
- 373. Detre JA, Wang J, Wang Z, Rao H. Arterial spin-labeled perfusion MRI in basic and clinical neuroscience. Curr Opin Neurol 2009;22:348-55.
- 374. Fidani P, De Ioris MA, Serra A, et al. A multimodal strategy based on surgery, radiotherapy, ICE regimen and high dose chemotherapy in atypical teratoid/rhabdoid tumours: a single institution experience. Journal of neuro-oncology 2009;92:177-83.
- 375. Fusar-Poli P, Howes O, Valli I, et al. Multimodal functional imaging investigation before and after the onset of psychosis. The international journal of neuropsychopharmacology / official scientific journal of the Collegium Internationale Neuropsychopharmacologicum (CINP) 2009;12:579-81.
- 376. Nitkunan A, Barrick TR, Charlton RA, Clark CA, Markus HS. Multimodal MRI in cerebral small vessel disease: its relationship with cognition and sensitivity to change over time. Stroke 2008;39:1999-2005.
- 377. Hoth KF, Nash J, Poppas A, Ellison KE, Paul RH, Cohen RA. Effects of cardiac resynchronization therapy on health-related quality of life in older adults with heart failure. Clinical interventions in aging 2008;3:553-60.
- 378. Cohen RA, Paul RH, Ott BR, et al. The relationship of subcortical MRI hyperintensities and brain volume to cognitive function in vascular dementia. J Int Neuropsychol Soc 2002;8:743-52.
- 379. Boyle PA, Paul RH, Moser DJ, Cohen RA. Executive impairments predict functional declines in vascular dementia. Clin Neuropsychol 2004;18:75-82.
- 380. Brickman AM, Zimmerman ME, Paul RH, et al. Regional white matter and neuropsychological functioning across the adult lifespan. Biol Psychiatry 2006;60:444-53.
- 381. Cohen RA, Browndyke JN, Moser DJ, Paul RH, Gordon N, Sweet L. Long-term citicoline (cytidine diphosphate choline) use in patients with vascular dementia: neuroimaging and neuropsychological outcomes. Cerebrovasc Dis 2003;16:199-204.
- 382. Garrett KD, Browndyke JN, Whelihan W, et al. The neuropsychological profile of vascular cognitive impairment--no dementia: comparisons to patients at risk for cerebrovascular disease and vascular dementia. Arch Clin Neuropsychol 2004;19:745-57.
- 383. Paul R, Moser D, Cohen R, Browndyke J, Zawacki T, Gordon N. Dementia severity and pattern of cognitive performance in vascular dementia. Appl Neuropsychol 2001;8:211-7.
- 384. Sweet LH, Paul RH, Cohen RA, et al. Neuroimaging correlates of dementia rating scale performance at baseline and 12-month follow-up among patients with vascular dementia. J Geriatr Psychiatry Neurol 2003;16:240-4.

- 385. Cohen RA, de la Monte S, Gongvatana A, et al. Plasma cytokine concentrations associated with HIV/hepatitis C coinfection are related to attention, executive and psychomotor functioning. J Neuroimmunol
- 2011;233:204-10.
- 386. Gunstad J, Spitznagel MB, Paul RH, et al. Body mass index and neuropsychological function in healthy children and adolescents. Appetite 2008;50:246-51.
- 387. Gunstad J, Paul RH, Cohen RA, et al. Relationship between body mass index and brain volume in healthy adults. Int J Neurosci 2008;118:1582-93.
- 388. Gunstad J, Paul RH, Spitznagel MB, et al. Exposure to early life trauma is associated with adult obesity. Psychiatry research 2006;142:31-7.
- 389. Hassenstab JJ, Sweet LH, Del Parigi A, et al. Cortical thickness of the cognitive control network in obesity and successful weight loss maintenance: a preliminary MRI study. Psychiatry research 2012;202:77-9.
- 390. Brown GG, Clark C, Liu TT. Measurement of cerebral perfusion with arterial spin labeling: Part 2. Applications. J Int Neuropsychol Soc 2007;13:526-38.
- 391. Brown GG, Eyler Zorrilla LT, Georgy B, Kindermann SS, Wong EC, Buxton RB. BOLD and perfusion response to finger-thumb apposition after acetazolamide administration: differential relationship to global perfusion. J Cereb Blood Flow Metab 2003;23:829-37.
- 392. Brown GG, Perthen JE, Liu TT, Buxton RB. A primer on functional magnetic resonance imaging. Neuropsychology review 2007;17:107-25.
- 393. Trahan DE, Larrabee GJ, Quintana JW. Visual recognition memory in normal adults and patients with unilateral vascular lesions. J Clin Exp Neuropsychol 1990;12:857-72.
- 394. Larrabee GJ, Trahan DE, Curtiss G. Construct validity of the Continuous Visual Memory Test. Arch Clin Neuropsychol 1992;7:395-405.
- 395. Paolo AM, Troster AI, Ryan JJ. Test-retest stability of the Continuous Visual Memory Test in elderly persons. Arch Clin Neuropsychol 1998;13:617-21.
- 396. Paolo AM, Troster AI, Ryan JJ. Continuous Visual Memory Test performance in healthy persons 60 to 94 years of age. Arch Clin Neuropsychol 1998;13:333-7.
- 397. Snitz BE, Roman DD, Beniak TE. Efficacy of the Continuous Visual Memory Test in lateralizing temporal lobe dysfunction in chronic complex-partial epilepsy. J Clin Exp Neuropsychol 1996;18:747-54.
- 398. Hall S, Pinkston SL, Szalda-Petree AC, Coronis AR. The performance of healthy older adults on the Continuous Visual Memory Test and the Visual-Motor Integration Test: preliminary findings. Journal of clinical psychology 1996;52:449-54.
- 399. Harker KT, Connolly JF. Assessment of visual working memory using event-related potentials. Clin Neurophysiol 2007:118:2479-88.
- 400. Banos JH, Dickson AL, Greer T. A computer-assisted administration of the Continuous Visual Memory Test. Clin Neuropsychol 2001;15:551-5.
- 401. Retzlaff PD, Morris GL. Event-related potentials during the Continuous Visual Memory Test. Journal of clinical psychology 1996;52:43-7.
- 402. Andrade KC, Pontes-Neto OM, Leite JP, Santos AC, Baffa O, de Araujo DB. Quantitative aspects of brain perfusion dynamic induced by BOLD fMRI. Arg Neuropsiguiatr 2006;64:895-8.
- 403. Leoni RF, Mazzeto-Betti KC, Andrade KC, de Araujo DB. Quantitative evaluation of hemodynamic response after hypercapnia among different brain territories by fMRI. Neuroimage 2008;41:1192-8.
- 404. Kim SG, Rostrup E, Larsson HB, Ogawa S, Paulson OB. Determination of relative CMRO2 from CBF and BOLD changes: significant increase of oxygen consumption rate during visual stimulation. Magn Reson Med 1999;41:1152-61.
- 405. Kastrup A, Kruger G, Glover GH, Neumann-Haefelin T, Moseley ME. Regional variability of cerebral blood oxygenation response to hypercapnia. Neuroimage 1999;10:675-81.
- 406. Posse S, Kemna LJ, Elghahwagi B, Wiese S, Kiselev VG. Effect of graded hypo- and hypercapnia on fMRI contrast in visual cortex: quantification of T(\*)(2) changes by multiecho EPI. Magn Reson Med 2001;46:264-71.

- 407. Provencher SW. Automatic quantitation of localized *in vivo* 1H spectra with LCModel. NMR Biomed 2001;14:260-4.
- 408. Cohen RA, Harezlak J, Gongvatana A, et al. Cerebral metabolite abnormalities in human immunodeficiency virus are associated with cortical and subcortical volumes. J Neurovirol 2010;16:435-44. 409. Gongvatana A, Harezlak J, Buchthal S, et al. Progressive cerebral injury in the setting of chronic HIV infection and antiretroviral therapy. J Neurovirol 2013.
- 410. Paul RH, Ernst T, Brickman AM, et al. Relative sensitivity of magnetic resonance spectroscopy and quantitative magnetic resonance imaging to cognitive function among nondemented individuals infected with HIV. J Int Neuropsychol Soc 2008;14:725-33.
- 411. Paul RH, Yiannoutsos CT, Miller EN, et al. Proton MRS and neuropsychological correlates in AIDS dementia complex: evidence of subcortical specificity. J Neuropsychiatry Clin Neurosci 2007;19:283-92.
- 412. Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet 1986;1:307-10.
- 413. Bland JM, Altman DG. Measuring agreement in method comparison studies. Stat Methods Med Res 1999;8:135-60.
- 414. Fischl B, Sereno MI, Dale AM. Cortical surface-based analysis. II: Inflation, flattening, and a surface-based coordinate system. Neuroimage 1999;9:195-207.
- 415. Fischl B, Sereno MI, Tootell RB, Dale AM. High-resolution intersubject averaging and a coordinate system for the cortical surface. Human brain mapping 1999;8:272-84.
- 416. Fischl B, Dale AM. Measuring the thickness of the human cerebral cortex from magnetic resonance images. Proceedings of the National Academy of Sciences of the United States of America 2000;97:11050-5.
- 417. Lezak M. Neuropsychological Assessment. 3rd ed. New York, New York: Oxford University Press; 1995.
- 418. Boyle PA, Paul R, Moser D, Zawacki T, Gordon N, Cohen R. Cognitive and neurologic predictors of functional impairment in vascular dementia. Am J Geriatr Psychiatry 2003;11:103-6.
- 419. Baecke JA, Burema J, Frijters JE. A short questionnaire for the measurement of habitual physical activity in epidemiological studies. The American journal of clinical nutrition 1982;36:936-42.
- 420. Richardson MT, Ainsworth BE, Wu HC, Jacobs DR, Jr., Leon AS. Ability of the Atherosclerosis Risk in Communities (ARIC)/Baecke Questionnaire to assess leisure-time physical activity. Int J Epidemiol 1995;24:685-93.
- 421. Philippaerts RM, Lefevre J, Delvaux K, et al. Associations between daily physical activity and physical fitness in Flemish males: A cross-sectional analysis. Am J Hum Biol 1999;11:587-97.
- 422. Philippaerts RM, Westerterp KR, Lefevre J. Doubly labelled water validation of three physical activity questionnaires. Int J Sports Med 1999;20:284-9.
- 423. Philippaerts RM, Lefevre J. Reliability and validity of three physical activity questionnaires in Flemish males. Am J Epidemiol 1998;147:982-90.
- 424. Westerterp KR. Assessment of physical activity level in relation to obesity: current evidence and research issues. Med Sci Sports Exerc 1999;31:S522-5.
- 425. Quan SF, Howard BV, Iber C, et al. The Sleep Heart Health Study: design, rationale, and methods. Sleep 1997;20:1077-85.
- 426. Broderick JE, Junghaenel DU, Schneider S, Pilosi JJ, Stone AA. Pittsburgh and Epworth Sleep Scale Items: Accuracy of Ratings Across Different Reporting Periods. Behav Sleep Med 2012.
- 427. Craig SE, Kohler M, Nicoll D, et al. Continuous positive airway pressure improves sleepiness but not calculated vascular risk in patients with minimally symptomatic obstructive sleep apnoea: the MOSAIC randomised controlled trial. Thorax 2012;67:1090-6.
- 428. Silva GE, Vana KD, Goodwin JL, Sherrill DL, Quan SF. Identification of patients with sleep disordered breathing: comparing the four-variable screening tool, STOP, STOP-Bang, and Epworth Sleepiness Scales. J Clin Sleep Med 2011;7:467-72.
- 429. Kraemer HC, Wilson GT, Fairburn CG, Agras WS. Mediators and moderators of treatment effects in randomized clinical trials. Archives of general psychiatry 2002;59:877-83.

- 430. MacKinnon DP, Lockwood CM, Hoffman JM, West SG, Sheets V. A comparison of methods to test mediation and other intervening variable effects. Psychological methods 2002;7:83-104.
- 431. MacKinnon D. Introduction to statistical mediation analysis. New York: Lawrence Erlbaum Assoc.; 2008.
- 432. Muthén L, Muthén BO. Mplus User's Guide. . 6th ed. Los Angeles, CA: . Muthén & Muthén; 1999-2010.
- 433. Cohen J. Statistical power analysis for behavioral sciences. 1988.
- 434. Hsieh F, Dlock D, Larsen M. A simple method of sample size calculation for linear and logistic regression. Stat Med 1998;17:1623-34.
- 435. Hshieh F, Lavori P. Sample size calculations for the Cox proportional hazards regression model with nonbinary covariates. Controlled Clincal Trials 2000;21(6):552-60.
- 436. Schoenfeld D, . Sample size formula for proportional hazards regression model. Biometrics 1983;39:499-503.
- 437. Dupont W, Plummer W. Power and sample size: Calculation of studies involving linear regression. Controlled Clincal Trials 1998;19:589-601.